## **Appendix 16.1.9 Documentation of Statistical Methods**

## **Appendix 16.1.9.1 Integrated Analysis Plan**

• Integrated Analysis Plan, Version 1.0 – 31 July 2018

## **Appendix 16.1.9.2 Statistical Outputs**

- Supporting Document for Table 15.4.3.1 The Mixed Procedure
- Supporting Document for Table 15.4.3.2 The Mixed Procedure
- Supporting Document for Table 15.4.3.3 The Mixed Procedure
- Supporting Document for Table 15.4.3.4 The Mixed Procedure
- Supporting Document for Table 15.4.3.5 The Mixed Procedure

## **Integrated Analysis Plan**

Clinical Study Protocol Identification No. MS200095-0028

Title

Open-Label, Parallel-Group Phase 1 Study to Investigate the Effect of Various Degrees of Hepatic Impairment on the Pharmacokinetics, Safety and Tolerability of the c-Met Kinase

Inhibitor Tepotinib

Study Phase

Ι

Investigational Medicinal

Tepotinib

Product(s)

Clinical Study Protocol

24 April 2018 / Version 2.0

Version

Integrated Analysis Plan Author Coordinating Author

Function

, Merck PI
Author(s) / Data Analyst(s)
, IQVIA PI

Integrated Analysis Plan Date and Version 31 July 2018 / Version 1.0

Integrated Analysis Plan Reviewers

| Function | Name |
|----------------------------|------|
| PI , IQVIA | PI |
| PI , IQVIA | PI |
| PI , IQVIA | PI |
| PI , IQVIA | PI |
| Medical Responsible, Merck | PI |
| PI , Merck | PI |
| PI , Merck | PI |
| PI , Merck | PI |
| PI , Merck | PI |
| PI , Merck | PI |
| PI , Merck | PI |
| PI , Merck | PI |

#### Confidential

This document is the property of Merck KGaA, Darmstadt, Germany, or one of its affiliated companies.

It is intended for restricted use only and may not - in full or part - be passed on, reproduced, published or used without express permission of Merck KGaA, Darmstadt, Germany or its affiliate.

Copyright © 2018 by Merck KGaA, Darmstadt, Germany or its affiliate. All rights reserved.

## Signature Page

Integrated Analysis Plan: MS200095-0028

Open-Label, Parallel-Group Phase 1 Study to Investigate the Effect of Various Degrees of Hepatic Impairment on the Pharmacokinetics, Safety and Tolerability of the c-Met Kinase Inhibitor Tepotinib

| Mercl | k responsible | Date | Signature |
|-------|---------------|-------------|--------------------|
| PI | , PI | Via ELDORAD | O approval process |
| PI | , PI | Via ELDORAD | O approval process |

## 1 Table of Contents

| Integrated Analys | sis Plan | 1 |
|---|---|---|
| Signature Page | | 2 |
| 1 | Table of Contents | 3 |
| 2 | List of Abbreviations and Definition of Terms | 5 |
| 3 | Modification History | 8 |
| 4 | Purpose of the Integrated Analysis Plan | 8 |
| 5 | Objectives and Endpoints | 8 |
| 6 | Overview of Planned Analyses | 9 |
| 6.1 | Interim Analysis | 9 |
| 6.2 | Final Analysis | 9 |
| 7 | Changes to the Planned Analyses in the Clinical Study Protocol | 9 |
| 8 | Protocol Deviations and Analysis Sets | 9 |
| 8.1 | Definition of Protocol Deviations | 9 |
| 8.2 | Definition of Analysis Sets and Subgroups | 10 |
| 9 | General Specifications for Data Analyses | 11 |
| 10 | Study Subjects | 12 |
| 10.1 | Disposition of Subjects and Discontinuations | 12 |
| 10.2 | Protocol Deviations | 13 |
| 10.2.1 | Important Protocol Deviations | 13 |
| 10.2.2 | Reasons Leading to the Exclusion from an Analysis Set | 13 |
| 11 | Demographics and Other Baseline Characteristics | 13 |
| 11.1 | Demographics | 13 |
| 11.2 | Medical History | 13 |
| 11.3 | Other Baseline Characteristics | 14 |
| 12 | Previous or Concomitant Medications/Procedures | 14 |
| 13 | Treatment Compliance and Exposure | 14 |
| 14 | Efficacy Analyses | 14 |
| 15 | Safety Analyses | 14 |
| 15.1 | Adverse Events | 14 |
| 15.1.1 | All Adverse Events | 15 |


 $I\,N\,F\,O\,R\,M\,A\,T\,I\,O\,N$ 

# Tepotinib (MSC2156119J) Tepotinib Hepatic Impairment Trial MS200095-0028

| 15.1.2 | Adverse Events Leading to Study Discontinuation | 15 |
|---|---|---|
| 15.2 | Deaths, Other Serious Adverse Events, and Other Significant Adverse Events | 16 |
| 15.2.1 | Deaths | 16 |
| 15.2.2 | Serious Adverse Events | 16 |
| 15.3 | Clinical Laboratory Evaluation. | 16 |
| 15.4 | Vital Signs | 16 |
| 15.5 | Other Safety or Tolerability Evaluations | 16 |
| 16 | Analyses of Other Endpoints | 17 |
| 16.1 | Pharmacokinetics | 17 |
| 16.1.1 | Primary Endpoints | 17 |
| 16.1.2 | Secondary Endpoints | 18 |
| 16.1.3 | Concentration Data | 19 |
| 16.1.4 | Estimation of Pharmacokinetic Parameters | 20 |
| 16.2 | Pharmacodynamics | 23 |
| 17 | References | 23 |
| 18 | Appendices | 23 |

#### 2 **List of Abbreviations and Definition of Terms**

**ADAM** Analysis Data Model

ΑE Adverse event

**ALBI** Albumin-Bilirubin **ANOVA** Analysis of variance

**AST** Aspartate aminotransferase

**AUC** Area under the plasma concentration-time curve

The AUC from time zero (dosing time) extrapolated to infinity  $AUC_{0-\infty}$ 

The AUC for unbound drug from time zero (dosing time) extrapolated to  $AUC_{0-\infty,u}$ 

infinity

 $AUC_{0-t}$ The AUC from time zero (dosing time) to the last sampling time ( $t_{last}$ ) at

which the concentration is at or above the lower limit of quantification

AUCextra% The AUC from time  $t_{last}$  extrapolated to infinity given as percentage of

 $AUC_{0-\infty}$ 

BLQ Below the lower limit of quantification

BMI Body mass index CI Confidence interval

CL/f The apparent total body clearance of drug following extravascular

administration.

CL/f<sub>.u</sub> The apparent total body clearance of unbound drug following

extravascular administration.

 $C_{max}$ Maximum observed plasma concentration

Maximum observed unbound plasma concentration  $C_{\text{max,u}}$ 

**CRF** Case report form

CSP Clinical study protocol **CSR** Clinical study report CV% Coefficient of variation

**ECG** Electrocardiogram

FSH Follicle-stimulating hormone

 $f_{n}$ Average free fraction of analyte, ie unbound

GCP Good Clinical Practice

GeoCV% Geometric coefficient of variation

6/88

## Tepotinib (MSC2156119J) Tepotinib Hepatic Impairment Trial MS200095-0028

GeoMean Geometric mean

IAP Integrated analysis plan

ICH International Council for Harmonisation

IMP Investigational medicinal product

LLOQ Lower limit of quantification

Max Maximum

Mean Arithmetic mean

MedDRA Medical Dictionary for Regulatory Activities

Min Minimum

 $\begin{array}{ll} \text{MRAUC}_{0\text{--}\infty} & \text{Metabolite to parent drug ratio for AUC}_{0\text{--}\infty} \\ \text{MRC}_{\text{max}} & \text{Metabolite to parent drug ratio for $C_{\text{max}}$} \end{array}$ 

MW Molecular weight

N, n Number of subjects or number of non-missing observations

NCI National Cancer Institute

NCI-CTCAE National Cancer Institute – Common Terminology Criteria for Adverse

**Events** 

ODWG Organ Dysfunction Working Group
PK Pharmacokinetic/Pharmacokinetics

PT Preferred Term
Q1 25th percentile
Q3 75th percentile

SAE Serious adverse event SD Standard deviation

SDTM Study Data Tabulation Model

SEM Standard error of the mean

SI Système International SOC System Organ Class

 $t_{1/2}$  Apparent terminal half-life

TEAE Treatment-emergent adverse event

t<sub>last</sub> The last sampling time at which the concentration is at or above the

lower limit of quantification

t<sub>max</sub> The time to reach the maximum observed concentration

## Tepotinib (MSC2156119J) Tepotinib Hepatic Impairment Trial MS200095-0028

ULN Upper limit of normal

Vz/F Apparent volume of distribution during the terminal phase following

extravascular administration

WHO DDE Enhanced World Health Organization Drug dictionary

 $\lambda_z$  Terminal elimination rate constant

## 3 Modification History

| Unique<br>Identifier for<br>Version | Date of<br>IAP Version | Aut | hor | Changes from the Previous Version |
|---|---|---|---|---|
| 1.0 | 31Jul2018 | PI | | Original document |
| | | PI | | |
| | | PI | | |

## 4 Purpose of the Integrated Analysis Plan

The purpose of this integrated analysis plan (IAP) is to document technical and detailed specifications for the final analysis of data collected for protocol MS200095-0028. Results of the analyses described in this IAP will be included in the clinical study report (CSR). Additionally, the planned analyses identified in this IAP will be included in regulatory submissions or future manuscripts. Any post-hoc or unplanned analyses performed to provide results for inclusion in the CSR but not identified in this prospective IAP will be clearly identified in the CSR.

The IAP is based upon the clinical study protocol (CSP) and is prepared in compliance with International Council for Harmonisation (ICH) E9. The first version (version 1.0) of this IAP focused on the detailed description of the statistical analyses for pharmacokinetics (PK) and safety variables. The Part 2 of the study is optional for which the analysis is not currently defined in this IAP.

## 5 Objectives and Endpoints

| | Objective | Endpoint | IAP<br>Section |
|---|---|---|---|
| Primary<br>Objective | To assess the PK of tepotinib in subjects with various degrees of impaired hepatic function (in comparison to healthy subjects) | Primary Endpoints • Tepotinib (plasma) area under the curve from time zero to the last quantifiable concentration sampling time (AUC <sub>D+</sub> ), area under the curve from time zero to infinity (AUC <sub>O-∞</sub> ), and maximum concentration observed (C <sub>max</sub> ) | 16.1 |
| Secondary<br>Objectives | To further investigate the PK of tepotinib and its metabolites MSC2571109 and MSC2571107 in subjects with various degrees of impaired hepatic function (in comparison to healthy subjects) | Secondary Endpoints Tepotinib (plasma) time to reach maximum plasma concentration (tmax), half-life (t1/2), apparent total body clearance (CL/f), apparent volume of distribution (Vz/f), the extrapolated part of AUC <sub>0-m</sub> (AUC <sub>extra%</sub> ); The free fraction (ie, unbound) of tepotinib will be determined to estimate unbound parameters AUC <sub>0-m</sub> , Cmax,u, and CL/f,u Tepotinib metabolites MSC2571109 and MSC2571107 (plasma), AUC <sub>0-t</sub> , AUC <sub>0-m</sub> , Cmax, tmax, t <sub>1/2</sub> , AUC <sub>extra%</sub> , and metabolite to parent drug ratio for AUC <sub>0-m</sub> (MRAUC <sub>0-m</sub> ) and metabolite to parent drug ratio for C <sub>max</sub> (MRC <sub>max</sub> ) | 16.1 |

| Objective | Endpoint | IAP<br>Section |
|---|---|---|
| To assess safety and tolerability of tepotinib in subjects with various degrees of impaired hepatic function (in comparison to healthy subjects). | Occurrence of treatment-emergent adverse<br>events (TEAEs), changes from baseline in<br>laboratory safety tests, 12-lead<br>electrocardiograms (ECG) morphology and time<br>intervals (PR, QRS, RR, QT, and QTcF), and vital<br>signs | 15 |

The analyses of the endpoints will be described in the respective sections for PK and safety, regardless of whether the endpoint is a primary endpoint or not.

## **6** Overview of Planned Analyses

## 6.1 Interim Analysis

There is no formal interim analysis planned.

## 6.2 Final Analysis

All final, planned analyses identified in the CSP and this IAP will be performed only after the last subject has completed the End of Study visit with all study data in-house, all data queries resolved, and the database locked.

A data review meeting will be held prior to database lock. In addition, no database can be locked until this IAP has been approved.

## 7 Changes to the Planned Analyses in the Clinical Study Protocol

There are no changes to the planned analyses.

## **8** Protocol Deviations and Analysis Sets

#### 8.1 Definition of Protocol Deviations

Important protocol deviations or events are protocol deviations or events that might significantly affect the completeness, accuracy, and/or reliability of the study data or that might significantly affect a subject's rights, safety, or well-being.

The following important deviations or events will be identified and confirmed prior to or at the Data Review Meeting:

- Subjects that are dosed on the study despite not satisfying the inclusion criteria
- Subjects that develop withdrawal criteria whilst on the study but are not withdrawn
- Subjects that receive an incorrect dose

- Subjects that receive a prohibited concomitant medication
- Deviation from Good Clinical Practice (GCP)
- Other events/factors related to PK data include, but may not be limited to, the following:
  - Sample processing errors that may lead to incorrect bioanalytical results
  - o Incomplete samples collected
  - o Use of prohibited medication that could affect PK
  - $\circ$  Events that could affect PK (ie such as vomiting within 2 times the median  $t_{max}$ , after dosing), to be evaluated on a case-by-case basis.

Subset of these important protocol deviations are considered clinically important, if leading to the exclusion of a subject from an analysis set (see Section 8.2).

All protocol deviations are documented in Study Data Tabulation Model (SDTM) datasets whether identified through site monitoring, medical review or programming.

## 8.2 Definition of Analysis Sets and Subgroups

#### **Screening Analysis Set**

The Screening Analysis Set will include all subjects who provide signed informed consent, regardless of treatment status in the study. This analysis set will be used for subject disposition.

#### Safety Analysis Set

The Safety Analysis Set will include all subjects who receive the study treatment. All safety analyses will be based on this analysis set.

#### **Pharmacokinetic Analysis Set**

The PK Analysis Set will include all subjects who receive the study treatment and have at least 1 postdose PK measurement without important protocol deviations/violations or events that may affect the PK. All PK analyses will be based on this analysis set.

The use of the analysis sets in the different analyses (no subgroup analyses are planned) is presented in the following table:

| Analyses | Screening<br>Analysis Set | Safety<br>Analysis Set | PK Analysis<br>Set |
|---|---|---|---|
| Subject Disposition | ✓ | | |
| Baseline Assessments | | ✓ | |
| Previous or Concomitant<br>Medications / Procedures | | ✓ | |
| Treatment Compliance and | | ✓ | |

| Analyses | Screening<br>Analysis Set | Safety<br>Analysis Set | PK Analysis<br>Set |
|---|---|---|---|
| Exposure | | | |
| PK Analysis | | | ✓ |
| Safety and Tolerability | | ✓ | |

#### **General Specifications for Data Analyses** 9

### Listings

All listings will be sorted by hepatic function group (impairment and healthy control), subject, and/or scheduled timepoint, as appropriate. Data from assessments which are only performed before administration of the investigational medicinal product (IMP) will be sorted by subject and scheduled timepoint (if appropriate).

#### **Tables**

All data will be summarized by hepatic function group and/or scheduled timepoint, as appropriate. Repeated and unscheduled measurements included in the listings will not be used for statistical analyses or summaries, unless the repeated measurement was performed due to unreliable values/technical reasons, eg, clotted samples.

### **Presentation of Continuous and Qualitative Variables for Safety**

Continuous variables will be summarized using descriptive statistics, ie, number of subjects (N), number of non-missing observations (n), arithmetic mean (Mean), standard deviation (SD), median, 25th Percentile - 75th Percentile (Q1 - Q3), minimum (Min) and maximum (Max).

Qualitative variables will be summarized by counts and percentages.

Unless otherwise stated, the calculation of proportions will be based on the number of subjects in the analysis set of interest. Therefore, counts of missing observations will be included in the denominator and presented as a separate category.

When the analysis refers only to certain visits, percentages will be based on the number of subjects still present in the study at that visit, unless otherwise specified.

Mean, Median, Q1, Q3, Min, and Max will have the same precision as the raw data included in the SDTM datasets for non-derived data. Standard deviation will be presented with one digit more than the mean. Derived data will be rounded to reasonable digits whereas maximal digits should be available in Analysis Data Model (ADaM) datasets then the similar precision definitions will be followed for descriptive statistics. Percentage will be reported using 1 decimal digit, if not otherwise specified.


 $I\,N\,F\,O\,R\,M\,A\,T\,I\,O\,N$ 

#### **Definition of Baseline**

If not otherwise specified, "baseline" refers to the last non-missing scheduled measurement prior to dosing, as appropriate. It will in general correspond to Day 1 predose for laboratory parameters, vital signs, and ECG data. However, if a subject is missing the baseline collection, the previous non-missing evaluation (as applicable) will become the baseline value. If no baseline or previous to baseline evaluations exist then the baseline value will be treated as missing.

#### **Common Calculations**

For quantitative measurements:

• Change from baseline: Value at Visit X – Baseline Value

#### **Definition of Duration**

Duration will be calculated by the difference of start and stop/end date + 1 if not otherwise specified.

#### **Conversion Factors**

The following conversion factors will be used to convert days into months or years: 1 month = 30.4375 days, 1 year = 365.25 days.

#### **Handling of Missing Data**

Unless otherwise specified, missing data will not be replaced. Handling of missing data for PK parameter calculations are discussed under Section 16.1.

#### **Software**

Pharmacokinetic parameters will be derived using noncompartmental methods with the validated computer program Phoenix<sup>®</sup> WinNonlin<sup>®</sup> 6.4 or higher (Certara, L.P., Princeton, New Jersey, USA), and/or SAS<sup>®</sup> Windows Version 9.4 or higher (Statistical Analysis System, SAS-Institute, Cary, North Carolina, USA). Pharmacokinetic figures will be developed using SAS<sup>®</sup>. All statistical analyses will be performed using SAS<sup>®</sup>.

## 10 Study Subjects

The subsections in this section include specifications for reporting subject disposition and treatment/study discontinuations. Additionally, procedures for reporting protocol deviations are provided.

## 10.1 Disposition of Subjects and Discontinuations

A summary table describing the number and percentage of subjects (as applicable) in each of the following disposition categories will be produced by hepatic function group and overall:

- Total number of subjects screened (ie, subjects who gave informed consent)
- Number of subjects treated (used as denominator for percentage calculation for the categories below)
- Number of subjects who completed the study
- Number of subjects who discontinued the study/treatment, with the reason of discontinuation.

Corresponding individual listings for study termination status and study entry (including screening failures) will be presented. Subjects discontinued the study/treatment will be listed with the corresponding reasons.

Summary of the number and percentage (as applicable) of subjects included in each analysis set (as described in Section 8.2) will be presented.

#### 10.2 Protocol Deviations

## **10.2.1 Important Protocol Deviations**

The listing of important protocol deviations will be provided.

### 10.2.2 Reasons Leading to the Exclusion from an Analysis Set

For subjects and/or individual concentration or parameter data excluded from the PK Analysis Set, the reasons for exclusion will be listed.

## 11 Demographics and Other Baseline Characteristics

Demographics and baseline characteristics will be presented for the Safety Analysis Set.

### 11.1 Demographics

Descriptive statistics will be presented for age, height, weight, and body mass index (BMI). Frequency counts and percentages will be presented for sex (gender), race, and ethnicity. The summary will be performed by hepatic function group and overall.

Subjects with hepatic impairment will be assigned to a group of mild (Child-Pugh class A) or moderate (Child-Pugh class B) hepatic impairment at Screening by use of the Child-Pugh system. A listing of points scored for observed findings based on Child-Pugh criteria will be presented.

## 11.2 Medical History

Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), current version, and listed. Prior surgery, if any, will also be listed.

#### 11.3 Other Baseline Characteristics

Other baseline characteristics and assessments, including nicotine and alcohol consumption, virus screen, alcohol breathalyzer test, cotinine test, drugs of abuse screen, pregnancy test in women, and follicle-stimulating hormone (FSH) in postmenopausal women, will be listed.

#### 12 Previous or Concomitant Medications/Procedures

Medications will be presented for the Safety Analysis Set.

Previous medications are defined as any medication discontinued prior to the IMP administration. Concomitant medications are defined as any medication taken during the course of the study, with a starting date greater than or equal to the IMP administration, or with a starting date prior to the IMP administration and ongoing at the time of the IMP administration.

The Enhanced World Health Organization Drug dictionary (WHO DDE), current version, will be used for coding of prior and concomitant medications.

Previous and concomitant medications, as well as concomitant procedures, if any, will be listed.

## 13 Treatment Compliance and Exposure

The IMP will be administered by the study center staff within the confines of the study center. The administration of IMP, meal consumption and fasting details will be listed for the Safety Analysis Set.

## 14 Efficacy Analyses

There are no efficacy endpoints and analyses defined for this CSP.

## 15 Safety Analyses

The subsections in this section include specifications for summarizing safety endpoints that are common across clinical studies such as adverse events (AEs), laboratory tests, and vital signs.

All analyses will be performed for the Safety Analysis Set.

#### 15.1 Adverse Events

All AEs recorded during the course of the study will be coded according to the MedDRA, current version, and each AE will be assigned to a System Organ Class (SOC) and a Preferred Term (PT).

Treatment-emergent AEs are those events with onset dates occurring after the IMP administration on Day 1. Any AE occurring before the IMP administration on Day 1 and resolved before the administration will be included in the AE listings, but will not be included in the summary tables (unless otherwise stated). These will be referred to as "pre-treatment".

In case of (partly) incomplete AE-related dates, the available information will be used in a conservative approach to determine whether the AE is treatment-emergent.

All analyses described in this section will be based on TEAEs if not otherwise specified.

#### 15.1.1 All Adverse Events

Treatment-emergent adverse events will be summarized by hepatic function group and overall in tables with:

- The number and percentage of subjects with any TEAE, any IMP related TEAE, any serious TEAE, any IMP related serious TEAE, any grade >=3 TEAE, any IMP related grade >=3 TEAE, any TEAE leading to death, any IMP related TEAE leading to death, any TEAE leading to study discontinuation
- The number and percentage of subjects with at least one TEAE by SOC and PT
- The number and percentage of subjects with at least one TEAE by SOC, PT, and worst grade according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), current version
- The number and percentage of subjects with at least one IMP related TEAE by SOC and PT
- The number and percentage of subjects with at least one TEAE by PT only, sorted in decreasing incidence overall
- The number and percentage of subjects with at least one non-serious TEAE by SOC and PT.

Unless otherwise stated, AEs will be displayed with SOC terms sorted alphabetically and PTs within each SOC term sorted in decreasing incidence overall.

For determining incidence counts, if a subject experiences more than one occurrence of the same TEAE, the subject will only be counted once for that TEAE.

If an AE is reported for a given subject more than once during treatment, the worst grade and the worst relationship to study treatment will be tabulated.

Adverse events related to IMP are those events with relationship missing or 'related'.

In case a subject had events with missing and non-missing grade, the maximum of the non-missing grade will be displayed.

## 15.1.2 Adverse Events Leading to Study Discontinuation

A listing of TEAEs leading to study discontinuation, if any, will be provided.

# 15.2 Deaths, Other Serious Adverse Events, and Other Significant Adverse Events

#### **15.2.1** Deaths

All deaths as well as reason for death will be based on information from the "Report of Subject Death" case report forms (CRFs). Listing of deaths, if any, will be provided displaying date and cause of death (including TEAE leading to death and relatedness to trial treatment, when applicable), and date and time of treatment administration.

#### 15.2.2 Serious Adverse Events

A listing of serious TEAEs, if any, will be provided.

## 15.3 Clinical Laboratory Evaluation

All clinical laboratory data will be stored in the database in the units in which they were reported with the laboratory reference ranges. Listings and summary statistics at each assessment time will be presented using the Système International (SI) units. Laboratory data not reported in SI units will be converted to SI units before processing.

Continuous clinical laboratory data (hematology and biochemistry) will be summarized by hepatic function group and timepoint using descriptive statistics for baseline (see definition in Section 9), each evaluation during the study, and change from baseline to each evaluation.

When applicable, laboratory results will be graded using the NCI-CTCAE, current version, and summarized by worst post-baseline toxicity grade and shift from baseline to highest grade.

Based upon laboratory normal ranges, these laboratory test results will be categorized according to the normal range as low (below the lower limit), normal (within the normal range), and high (above the upper limit). Listings of all clinical laboratory data for each subject will be provided with values outside the normal ranges indicated. Listings of abnormal test results (low and high) will be provided.

## 15.4 Vital Signs

Vital signs data (including oral temperature, systolic and diastolic blood pressure, and pulse rate) will be summarized by hepatic function group and timepoint using descriptive statistics for baseline (see definition in Section 9), each evaluation during the study, and change from baseline to each evaluation. Listing of vital signs data will be provided.

## 15.5 Other Safety or Tolerability Evaluations

Safety 12-lead ECG data will be summarized by hepatic function group and time point using descriptive statistics for baseline (see definition in Section 9), each evaluation during the study, and change from baseline to each evaluation. Listings of ECG data will be provided. Overall


INFORMATION

ECG assessments (normal, abnormal/not clinically significant, abnormal/clinically significant) will also be listed.

Clinically significant, abnormal findings from the physical examination are to be reported as AEs. Separate summary or listing of the physical examination will not be provided.

## 16 Analyses of Other Endpoints

#### 16.1 Pharmacokinetics

All statistical analyses and descriptive summaries of PK data will be performed on the PK Analysis Set. Pharmacokinetic parameters will not be summarized if more than 50% of the dataset are missing for a respective parameter.

## **16.1.1 Primary Endpoints**

As the primary analysis, an analysis of variance (ANOVA) model including hepatic function group as a fixed effect will be applied to log-transformed tepotinib PK parameters  $AUC_{0-t}$ ,  $AUC_{0-\infty}$ , and  $C_{max}$  of the subjects with Mild Impairment (Child-Pugh class A), Moderate Impairment (Child-Pugh class B) and the healthy subjects of the matched control group. Least-squares means and corresponding 95% CIs by group, differences and corresponding 90% CIs between the hepatic impairment groups and control will be estimated on the log scale. Point estimates and CIs will be back-transformed to the original scale for presentation.

Additionally, a generalized linear model including hepatic function group and sex (gender) as fixed effects, age and weight as covariates, will be applied to the same primary PK parameters.

Boxplots will be prepared for AUC<sub>0-t</sub>, AUC<sub>0- $\infty$ </sub> and C<sub>max</sub> of tepotinib by hepatic function group.

Primary endpoints will be descriptively summarized as described below for secondary endpoints.

In a further analysis, the subjects with liver impairment will be evaluated according to the Albumin-Bilirubin (ALBI) score and the Organ Dysfunction Working Group (ODWG) classification (1, 2).

To categorize subjects based on the ALBI score (1), the following equation will be used: linear predictor = (log10(bilirubin)  $\times$  0.66) + (albumin  $\times$  -0.085), where bilirubin is in  $\mu$ mol/L and albumin in g/L. Calculating the subject-level linear prediction (xb) and applying the cut points assigned each subject to one of three prognostic groups, named the ALBI grade, 1 to 3. The cut points are as follows: xb  $\leq$  -2.60 (ALBI grade 1), more than -2.60 to  $\leq$  -1.39 (ALBI grade 2), and xb more than -1.39 (ALBI grade 3). The linear prediction values will be derived for healthy subjects as well.

To categorize subjects based on the ODWG classification (2), the following will be followed: subjects will be assigned to four groups based on hepatic function, defined according to bilirubin and aspartate aminotransferase (AST) levels relative to the upper limit of normal (ULN) using the classification developed for organ dysfunction studies by the National Cancer Institute (NCI)

ODWG. Normal function is defined as bilirubin and AST  $\leq$ ULN. Subjects with mild hepatic impairment have bilirubin  $\leq$ ULN and AST >ULN, or bilirubin >1.0–1.5 x ULN (with any AST). Moderate and severe hepatic impairments are defined as bilirubin >1.5–3 x ULN and >3 x ULN, respectively, with any AST.

The classifications for both ALBI and ODWG will be derived using the laboratory data obtained at Screening, while the same will be performed for laboratory data at Day 1 predose, for comparison purpose. These additional classifications will be presented in a listing.

Using the ALBI or ODWG classification, the generalized linear model including hepatic function group and sex (gender) as fixed effects, age and weight as covariates, will be applied to the same primary PK parameters. In addition, a similar model using the ALBI linear prediction values as a continuous variable, will also be performed.

## **16.1.2** Secondary Endpoints

Secondary endpoints are: Tepotinib (plasma)  $t_{max}$ ,  $t_{1/2}$ , CL/f, Vz/f,  $AUC_{extra\%}$ ; unbound tepotinib parameters  $AUC_{0-\infty,u}$ ,  $C_{max,u}$ , and  $CL/f_{,u}$ 

Tepotinib metabolites MSC2571109 and MSC2571107 (plasma), AUC<sub>0-t</sub>, AUC<sub>0-∞</sub>, C<sub>max</sub>, t<sub>max</sub>, t<sub>1/2</sub>, AUC<sub>extra%</sub>, MRAUC<sub>0-∞</sub>, and MRC<sub>max</sub>.

All pharmacokinetic parameters data will be descriptively summarized using (refer to Section 9): n, Mean, SD, standard error of the mean (SEM), coefficient of variation (CV%), Min, Median, Max, Q1 and Q3 as appropriate, geometric mean (GeoMean), the geometric coefficient of variation (GeoCV%), and the 95% confidence interval (CI) for the GeoMean (LCI 95% GM, UCI 95% GM).

Non-derived data will have the same precision as SDTM data (number of digits) for the following descriptive statistics: mean, median, Q1, Q3, Min, and Max. Statistics on derived data (i.e., SD) is to be presented with one digit more than the mean.

PK parameter  $C_{max}$  will be reported with the same precision as the source data and mean  $t_{max}$  (h) will be reported to two decimal places. All other PK parameters will be reported to 3 significant figures. Descriptive statistics of PK parameter data will be calculated using full precision values, and rounded for reporting purposes only.

The following conventions will be applied when reporting individual values and descriptive statistics of PK parameter data:

Listings: 3 significant digits

Mean, Min, Median, Max, GeoMean, 95% CI, Q1 and Q3: 3 significant digits

SD, SEM: 4 significant digits

CV%, GeoCV%: 1 decimal place

For the secondary PK parameters  $AUC_{0-t}$ ,  $AUC_{0-\infty}$ , and  $C_{max}$  of the tepotinib metabolites, the primary ANOVA model including hepatic function group as a fixed effect as defined for the primary endpoints will be applied. Boxplots will also be provided as described for primary PK parameters included in the statistical analysis.

#### 16.1.3 Concentration Data

A listing of PK blood sample collection times by individual, as well as derived sampling time and time deviations, will be provided. Actual elapsed sample collection times will be rounded to two decimal places with units of hours. All PK concentrations will be reported and analyzed with the same precision as the source data provided by the bioanalytical laboratory or clinical laboratory regardless of how many significant figures or decimal places the data carry. Pharmacokinetic parameters and actual elapsed sample collection times will be rounded for reporting purposes in by-subject listings.

Plasma concentrations of tepotinib, its metabolites (MSC2571109 and MSC2571107) and the free-fraction of tepotinib in plasma will be listed and presented in summary tables by hepatic function group and/or nominal timepoint, as appropriate, showing: number of non-missing observations (n), Mean, SD, CV%, Min, median, and Max. Values below the lower limit of quantitation (LLOQ) will be identified as (BLQ), will be taken as zero for descriptive statistics. All data will be evaluated as observed; no imputation method for missing values will be used.

Descriptive statistics of PK concentration data will be calculated using values with the same precision as the source data, and rounded for reporting purposes only. The following conventions will be applied when reporting individual values and descriptive statistics of PK concentration data:

Listings: 3 significant digits

Mean, Min, Median, Max: 3 significant digits

SD: 4 significant digits

CV%: 1 decimal place

Pharmacokinetic plasma concentrations which are erroneous due to a protocol deviation (as defined in the protocol), documented handling error or analytical error (as documented in the bioanalytical report) may be qualified as invalid if agreed with the Sponsor prior to performing a statistical analysis. In this case the rationale must be provided in the CSR. Invalid concentrations will be flagged within the listings. Any other PK concentrations that appear implausible to the Pharmacokineticist/PK Data Analyst must not be excluded from the analysis. Any implausible data will be documented in the CSR.

Arithmetic mean plasma tepotinib (including free fraction tepotinib) and its metabolites (MSC2571109 and MSC2571107) concentration versus scheduled (nominal) time plots for all hepatic function groups will be provided using a linear and semi-logarithmic scale. Mean plots

will include SD bars (±SD) when plotted on a linear scale. The mean plasma concentration-time profiles will be plotted for subjects included in the PK Analysis Set.

Individual plasma tepotinib and its metabolites (MSC2571109 and MSC2571107) concentration versus actual time plots will be provided using a linear and semi-logarithmic scale. Plots of individual profiles of plasma tepotinib and its metabolites (MSC2571109 and MSC2571107) concentration versus actual time for all subjects within each hepatic function group, presented on a single plot (ie, spaghetti plots), will be provided by hepatic function group, separately, using a linear and semi-logarithmic scale.

#### 16.1.4 Estimation of Pharmacokinetic Parameters

For PK parameters, the standard rounding procedure will be as follows: in export datasets, as well as in the SDTM PP domain, PK parameters will be provided with full precision, and will not be rounded.

For the PK analysis, predose and postdose sample concentrations that are BLQ will be assigned a numerical value of zero for the calculation of PK parameters.

Predose samples that occur before the first drug administration will be assigned a time of 0 hour, as if the sample had been taken simultaneously with the IMP administration.

Pharmacokinetic parameters will be calculated using standard non-compartmental methods. Pharmacokinetic parameters will be evaluated and listed for all subjects who provide sufficient concentration-time data. At least 3 quantifiable, postdose concentration points will be required in the PK profile to obtain any PK parameter estimate.

Pharmacokinetic parameters will be calculated using the actual elapsed time since dosing, given with a precision of 14 significant digits or the SAS format Best12. In cases where the actual sampling time is missing, calculations will be performed using the scheduled time. Otherwise, there will be no further imputation of missing data other than for a missing predose concentration as stated above.

For each subject in the PK Analysis Set, the following PK parameters will be calculated for tepotinib and tepotinib metabolites MSC2571109 and MSC2571107, where appropriate:

| Symbol | Definition |
|---|---|
| AUC <sub>0-t</sub> | The AUC from time zero (= dosing time) to the last sampling time (t <sub>last</sub> ) at which the concentration is at or above the LLOQ. Calculated using the mixed log linear trapezoidal rule (linear up, log down). Units: ng x h/mL. |
| AUC <sub>0-∞</sub> | The AUC from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at $t_{last}$ , as estimated using the linear regression from $\lambda_z$ determination. AUC <sub>0-∞_pred</sub> =AUC <sub>0-t</sub> +C <sub>lastpred</sub> / $\lambda_z$ . |

| Symbol | Definition |
|---|---|
| | Units: ng x h/mL. |
| AUCextra% | The AUC from time $t_{last}$ extrapolated to infinity given as percentage of $AUC_{0\to\infty}$ . $AUC_{extra\%}$ = (extrapolated area/AUC <sub>0→∞</sub> ) *100. The predicted $AUC_{0\to\infty}$ should be used. Units: %. |
| CL/f | The apparent total body clearance of drug following extravascular administration. (tepotinib only) $CL/f = Dose_{p.o.}/AUC_{0-\infty\_pred}$ . Units: L/h. |
| C <sub>max</sub> | Maximum observed concentration, taken directly from the observed concentration-time profile. Units: ng/mL. |
| t <sub>max</sub> | The time to reach the maximum observed concentration collected during a dosing interval (unless otherwise defined, the first occurrence in case of multiple/identical $C_{max}$ values will be used). Units: h. |
| t <sub>1/2</sub> | Apparent terminal half-life. $t_{1/2} = \ln (2)/\lambda_{z}$ . Units: h. |
| Vz/f | The apparent volume of distribution during the terminal phase following extravascular administration $Vz/F = Dose/(AUC_{0-\infty\_pred} \times \lambda_z)$ following single dose. (tepotinib only). Units: L. |
| $\lambda_z$ | Terminal elimination rate constant (lambda_z). Determined from the terminal slope of the log-transformed concentration curve using linear regression on terminal data points of the curve. Units: h <sup>-1</sup> . |
| MRAUC <sub>0-∞</sub> | Metabolite (MSC2571109 or MSC2571107) $AUC_{0-\infty\_pred}$ to tepotinib $AUC_{0-\infty\_pred}$ ratio. |
| MRC <sub>max</sub> | Metabolite (MSC2571109 or MSC2571107) C <sub>max</sub> to tepotinib C <sub>max</sub> ratio. |

| Symbol | Definition |
|---|---|
| fu | Fraction of analyte unbound. Free fraction will be calculated as the ratio of free concentration divided by total concentration at a given sampling point. Both unbound (ie, plasma ultrafiltrate) concentrations and unbound fractions will be listed for each scheduled sample collection. The average $f_u$ will represent the average of all available fractions (assuming concentration independent protein binding). If only a single unbound concentration is available, the derived fraction of the single timepoint for the respective analyte will be used for all calculations. If the unbound concentration is below the LLOQ at a given timepoint, that timepoint will be omitted from the calculation of the average and only the available timepoints will be used. If the unbound concentration falls below LLOQ in all 4 samples, $f_u$ and unbound PK parameters will not be presented. (tepotinib only) |
| C <sub>max,u</sub> | Maximum unbound plasma drug concentration, calculated as $C_{max}*f_u$ (tepotinib only) |
| AUC <sub>0-∞</sub> , <sub>u</sub> | Area under the concentration-time curve for unbound drug from time zero to infinity, calculated as $AUC_{0-\infty\_pred}$ *fu (or $AUC0$ -t*fu if $AUC_{0-\infty\_pred}$ is not adequately estimable (tepotinib only); |
| CL/f,u | Unbound apparent oral clearance, calculated as $CL/f_{,u} = Dose_{p.o.}/AUC_{0-\infty\_pred}/f_u$ (tepotinib only). Units: L/h |
| Note: Predicted will be presented | estimates for AUC <sub>0-∞</sub> , and all parameters derived (ie, AUC <sub>extrap</sub> %, AUC <sub>0-∞</sub> , <sub>u</sub> CL/f, CL/f, <sub>u</sub> , and Vz/F) |

If f<sub>u</sub> appears to be concentration dependent or time dependent, an alternate approach for calculation of unbound PK parameters may be employed and will be discussed in the CSR.

The following PK parameters will be calculated for diagnostic purposes and listed, but will not be summarized:

- The time interval (h) of the log-linear regression ( $\lambda_{z \text{ lower}}$ ,  $\lambda_{z \text{ upper}}$ ) to determine  $\lambda_{z}$
- Number of data points  $(N_{\lambda})$  included in the log-linear regression analysis to determine  $\lambda_z$
- Goodness-of-fit statistic (Rsq) for calculation of  $\lambda_z$
- The AUC from time  $t_{last}$  extrapolated to infinity given as percentage of AUC<sub>0-\infty</sub>. Units: \%.

The regression analysis for the terminal phase should contain data from at least 3 different timepoints consistent with the assessment of a straight line on the log-transformed scale. Phoenix WinNonlin best fit methodology will be used as standard. However, the PK scientist may adjust the regression analysis, if warranted by the data. The last quantifiable concentration should always be included in the regression analysis, while the concentration at t<sub>max</sub> and any concentrations < LLOQ which occur after the last quantifiable data point should not be used.

The Rsq should be  $\geq$  0.800, or AUC<sub>extra%</sub>  $\leq$  20.0%. If these criteria are not met, then the rate constants and all derived parameters (eg, AUC<sub>0- $\infty$ </sub>, AUC<sub>extra%</sub>, CL/f,  $\lambda_z$ , MRAUC<sub>0- $\infty$ </sub>, MRC<sub>max</sub>, t<sub>1/2</sub>, V<sub>z</sub>/f) will be included in the parameter output Listings and flagged as invalid for descriptive statistics. These exclusions are to be discussed appropriately. Any flags should be included in the study specific SDTM.

The IMP dose administered is given for the monohydrate hydrochloride salt (ie, 500 mg IMP). A conversion factor for the freebase IMP was calculated and will be applied when 'dose' is used in deriving PK parameter formulas needing a dose value (CL/f).

Conversion factor = Molecular weight (MW) of base IMP divided by MW of salt form IMP

492.574 g/mol / 547.05 g/mol = 0.9004 = conversion factor

Amount of dose \* conversion factor = actual dose of IMP: 500 mg \* 0.900 = 450 mg

No MW conversion factor for the parent-to-metabolite ratios will be applied.

A Phoenix WinNonlin NCA Core Output will be provided in a separate listing. Individual PK parameters will be calculated using actual sampling times.

Missing concentrations (eg, no sample, insufficient sample volume for analysis, no result, or result not valid) will be reported and displayed generally as "N.R.".

## 16.2 Pharmacodynamics

There are no pharmacodynamic assessments planned

#### 17 References

- 1. Johnson PJ, Berhane S, Kagebayashi C, et al. Assessment of liver function in patients with hepatocellular carcinoma: a new evidence-based approach-the ALBI grade. *J Clin Oncol*. 2015; 33(6) 550-558.
- LoRusso PM, Venkatakrishnan K, Ramanathan RK, et al. Pharmacokinetics and safety of bortezomib in patients with advanced malignancies and varying degrees of liver dysfunction: Phase 1 NCI Organ Dysfunction Working Group study NCI-6432. *Clin Cancer Res.* 2012; 18(10), doi:10.1158/1078-0432.CCR-11-2873.

## **Appendices**

There are no appendices.

## CTP MS200095-0028 Integrated Analysis Plan Version 1

## **ELECTRONIC SIGNATURES**

| Sig | gned by | Meaning of Signature | Server Date<br>(dd-MMM-yyyy HH:mm 'GMT'Z) |
|---|---|---|---|
| PI | | Business Approval | 02-Aug-2018 12:37 GMT+02 |
| PI | | Technical Approval | 06-Aug-2018 10:23 GMT+02 |

Supporting Document for Tables 15.4.3.1.1/2, 15.4.3.6.1/2, and 15.4.3.7.1/2

The Mixed Procedure

ANAL=Primary Model ANALYTEN=1 ANALYTE=Tepotinib PARM=AUC0-t (ng\*h/mL) PARAMCD=AUCLST

| Model Information | no |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| el<br>on | Values | 1 2 3 |
|----------------------------|--------|-------|
| Class Level<br>Information | Levels | 3 |
| υĤ | Class | GRP |

| | 1 | 4 | 0 | 1 | 18 |
|---|---|---|---|---|---|
| Dimensions | Covariance Parameters | Columns in X | Columns in Z | Subjects | Max Obs per Subject |

| Number of Observations | |
|-----------------------------|----|
| Number of Observations Read | 18 |
| Number of Observations Used | 18 |

Number of Observations

Number of Observations Not Used

0

| covariance<br>Parameter<br>Estimates | Estimate | 0.1497 |
|--------------------------------------|----------|----------|
| Covar<br>Paran<br>Estin | Cov Parm | Residual |

| Fit Statistics | |
|--------------------------|------|
| -2 Res Log Likelihood | 19.5 |
| AIC (Smaller is Better) | 21.5 |
| AICC (Smaller is Better) | 21.8 |
| BIC (Smaller is Better) | 22.2 |

| | | Ω | Solution for Fixed Effects | or F | ixed Effe | cts | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Actual<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Intercept | | 10.0665 | 0.1580 15 | 15 | 63.73 | | 0.05 | <.0001 0.05 9.7298 10.4032 | 10.4032 |
| GRP | 1 | 0.1370 | 0.1370 0.2234 15 | 15 | | 0.61 0.5489 0.05 -0.3391 0.6132 | 0.05 | -0.3391 | 0.6132 |
| GRP | 2 | 0.08370 | 0.08370 0.2234 15 | 15 | 0.37 | 0.37 0.7131 0.05 -0.3924 0.5599 | 0.05 | -0.3924 | 0.5599 |
| GRP | 3 | 0 | | | | | | | |

| ffects | Pr > F | 0.8280 |
|---------|-----------|--------|
| Fixed E | F Value | 0.19 |
| ts of | Den<br>DF | 15 |
| Tes | Num<br>DF | 2 |
| Type 3 | Effect | GRP |

| | | EST. | Estimates | tes | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Standard | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Mild vs Healthy | -0.05331 | 0.2234 15 | 15 | -0.24 | 0.8146 | | 0.1 -0.4449 0.3383 | 0.3383 |
| Moderate vs Healthy | -0.1370 | 0.2234 15 | 15 | -0.61 | 0.5489 | | 0.1 -0.5286 0.2546 | 0.2546 |

| | | | Least | Sque | Least Squares Means | τΩ | | | |
|---|---|---|---|---|---|---|---|---|---|
| Act<br>Tre<br>Effect (N) | Actual<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | ndard | Alpha | Lower | Upper |
| GRP | 1 | 10.2035 | 10.2035 0.1580 15 | 15 | 64.59 | < .0001 | 0.05 | 9.8668 | <.0001 0.05 9.8668 10.5402 |
| GRP | 2 | 10.1502 | 0.1580 15 | 15 | 64.26 | | 0.05 | 9.8135 | <.0001 0.05 9.8135 10.4869 |
| GRP | 3 | 10.0665 | 0.1580 15 | 15 | 63.73 | | 0.05 | 9.7298 | <.0001 0.05 9.7298 10.4032 |

Supporting Document for Tables 15.4.3.1.1/2, 15.4.3.6.1/2, and 15.4.3.7.1/2

The Mixed Procedure

ANAL=Primary Model ANALYTEN=1 ANALYTE=Tepotinib PARM=AUC0-inf (ng\*h/mL) PARAMCD=AUCIFP

| Model Information | n |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| el<br>on | Values | 123 |
|----------------------------|--------|-----|
| Class Level<br>Information | Levels | ε |
| ט ה | Class | GRP |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | Τ |
| Columns in X | 4 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 18 |

| Number | οĘ | Observations | |
|-----------------|--------------|--------------|----|
| Number of Obser | Observations | Read | 18 |
| Number of Obser | Observations | Used | 18 |

Number of Observations
Number of Observations Not Used 0

| Covariance<br>Parameter<br>Estimates | Estimate | 0.1434 |
|--------------------------------------|----------|----------|
| Covar<br>Paran<br>Estin | Cov Parm | Residual |

| Fit Statistics | |
|--------------------------|------|
| -2 Res Log Likelihood | 18.8 |
| AIC (Smaller is Better) | 20.8 |
| AICC (Smaller is Better) | 21.1 |
| BIC (Smaller is Better) | 21.5 |

| | | Ø | Solution for Fixed Effects | or F | ixed Effe | cts | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Actual<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Intercept | | 10.0921 | 0.1546 15 | 15 | 65.29 | | 0.05 | <.0001 0.05 9.7626 10.4216 | 10.4216 |
| GRP | 1 | 0.1287 | 0.1287 0.2186 15 | 15 | | 0.59 0.5647 0.05 -0.3372 0.5947 | 0.05 | -0.3372 | 0.5947 |
| GRP | 2 | 0.07732 | 0.2186 15 | 15 | 0.35 | 0.35 0.7285 0.05 -0.3886 0.5433 | 0.05 | -0.3886 | 0.5433 |
| GRP | 3 | 0 | | | | | | | |

| ffects | Pr > F | 0.8406 |
|---------|-----------|--------|
| Fixed E | F Value | 0.18 |
| ts of | Den<br>DF | 15 |
| Test | Num<br>DF | 2 |
| Type 3 | Effect | GRP |

| | | Est | Estimates | tes | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Standard | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Mild vs Healthy | -0.05141 | 0.2186 15 | 15 | -0.24 | 0.8173 | | 0.1 -0.4347 0.3318 | 0.3318 |
| Moderate vs Healthy | -0.1287 | 0.2186 15 | 15 | -0.59 | 0.5647 | | 0.1 -0.5120 0.2545 | 0.2545 |

| | | | Least | Sque | Least Squares Means | TO. | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Actual<br>Treatment (N) | Estimate | Standard<br>Error | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha Lower | Alpha | Lower | Upper |
| GRP | 1 | 10.2208 | 0.1546 15 | 15 | 66.12 | | 0.05 | 9.8913 | <.0001 0.05 9.8913 10.5503 |
| GRP | 2 | 10.1694 | 10.1694 0.1546 15 | 15 | 62.79 | | 0.05 | 9.8399 | <.0001 0.05 9.8399 10.4989 |
| GRP | 3 | 10.0921 | 10.0921 0.1546 15 | 15 | 65.29 | | 0.05 | 9.7626 | <.0001 0.05 9.7626 10.4216 |

32/88

Supporting Document for Tables 15.4.3.1.1/2, 15.4.3.6.1/2, and 15.4.3.7.1/2

The Mixed Procedure

ANAL=Primary Model ANALYTEN=1 ANALYTE=Tepotinib PARM=Cmax (ng/mL) PARAMCD=CMAX

| Model Information | no |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| el | Values | 123 |
|----------------------------|--------|-----|
| Class Level<br>Information | Levels | 3 |
| ט בו | Class | GRP |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | 1 |
| Columns in X | 4 |
| Columns in Z | 0 |
| Subjects | Τ |
| Max Obs per Subject | 18 |

| | 0 |
|---------------|--------------|
| rations | Used |
| rvat | Not |
| of Observa | ions |
| U | vat: |
| <b>lumber</b> | Observations |
| 7 | of |
| | Number |

| covariance<br>Parameter<br>Estimates | Estimate | 0.05441 |
|--------------------------------------|----------|----------|
| Covar<br>Parar<br>Estin | Cov Parm | Residual |

| Fit Statistics | |
|--------------------------|-----|
| -2 Res Log Likelihood | 4.3 |
| AIC (Smaller is Better) | 6.3 |
| AICC (Smaller is Better) | 9.9 |
| BIC (Smaller is Better) | 7.0 |

| | | SS | Solution for Fixed Effects | r Fi | xed Effe | cts | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Actual<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | | Lower Upper |
| Intercept | | 5.6642 | 5.6642 0.09523 15 | 15 | 59.48 | <.0001 | 0.05 | <.0001 0.05 5.4612 5.8671 | 5.8671 |
| GRP | 1 | 0.3423 | 0.3423 0.1347 15 | 15 | 2.54 | 2.54 0.0226 0.05 0.05523 0.6293 | 0.05 | 0.05523 | 0.6293 |
| GRP | 2 | 0.3664 | 0.1347 15 | 15 | 2.72 | 0.0158 0.05 0.07940 0.6535 | 0.05 | 0.07940 | 0.6535 |
| GRP | 3 | 0 | | | | | | | |

Type 3 Tests of Fixed Effects

Num Den F Value Pr > F

GRP 2 15 4.63 0.0271

| | | 田 | time | Estimates | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Standard | DF | t Value | ndard Error DF t Value Pr > t Alpha | Alpha | Lower | Lower Upper |
| Mild vs Healthy | 0.02417 | 0.1347 15 | 15 | 0.18 | 0.18 0.8599 | | 0.1 -0.2119 0.2603 | 0.2603 |
| Moderate vs Healthy -0.3423 0.1347 15 | -0.3423 | 0.1347 | 15 | | -2.54 0.0226 0.1 -0.5784 -0.1062 | 0.1 | -0.5784 | -0.1062 |

| | | | Least 2 | gdna | Least Squares Means | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Act<br>Tre<br>Effect (N) | Actual<br>Treatment (N) | Estimate | Standard<br>Error | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | | Lower Upper |
| GRP | 1 | 6.0064 | 6.0064 0.09523 15 | 15 | 80.69 | | 0.05 | <.0001 0.05 5.8035 6.2094 | 6.2094 |
| GRP | 2 | 9080.9 | 6.0306 0.09523 15 63.33 | 15 | 63.33 | | 0.05 | <.0001 0.05 5.8276 6.2336 | 6.2336 |
| GRP | 3 | 5.6642 | 5.6642 0.09523 15 | 15 | 59.48 | 1000.> | 0.05 | <.0001 0.05 5.4612 5.8671 | 5.8671 |

Supporting Document for Tables 15.4.3.1.1/2, 15.4.3.6.1/2, and 15.4.3.7.1/2

The Mixed Procedure

ANAL=Primary Model ANALYTEN=2 ANALYTE=Metabolite 2571107A PARM=AUCO-t (ng\*h/mL) PARAMCD=AUCLST

| Model Information | no |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| el<br>on | Values | 123 |
|----------------------------|--------|-----|
| Class Level<br>Information | Levels | 3 |
| D H | Class | GRP |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | Н |
| Columns in X | 4 |
| Columns in Z | 0 |
| Subjects | Τ |
| Max Obs per Subject | 18 |

| | Z | Number of Obse | of Observations | |
|-----------|----|----------------|-----------------|----|
| Number of | of | Observations | Read | 18 |
| $_{ m N}$ | of | Observations | Used | 18 |

| 0 | Used | Not | tions | Observations | of | Jumber |
|---|-------------|------|-------|--------------|----|--------|
| | bservations | rvat | 0 | nmber of | Z | |

| | (1) | 10 |
|--------------------------------------|----------|----------|
| Covariance<br>Parameter<br>Estimates | Estimate | 0.3645 |
| Covar<br>Parar<br>Estir | Cov Parm | Residual |

| | | S | Solution for Fixed Effects | r Fi | xed Effe | cts | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Actual<br>Treatment<br>(N) | Estimate | Standard | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | | Lower Upper |
| Intercept | | 8096.9 | 0.2465 15 | 15 | 28.24 | <.0001 | 0.05 | <.0001 0.05 6.4354 7.4861 | 7.4861 |
| GRP | 1 | 0.05676 | 0.05676 0.3486 15 | 15 | | 0.16 0.8728 0.05 -0.6862 0.7997 | 0.05 | -0.6862 | 0.7997 |
| GRP | 2 | 0.06146 | 0.3486 15 | 15 | 0.18 | 0.18 0.8624 0.05 -0.6815 0.8044 | 0.05 | -0.6815 | 0.8044 |
| GRP | 3 | 0 | | | | | | | |

Type 3 Tests of Fixed Effects

| Num Den | F Value | Pr > F GRP | 2 | 15 | 0.02 | 0.9809
| | | Est | Estimates | tes | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Standard | DF | t Value | undard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Mild vs Healthy | 0.004702 | 0.3486 15 | 15 | 0.01 | 0.9894 | 0.1 | 0.1 -0.6063 0.6158 | 0.6158 |
| Moderate vs Healthy -0.05676 | -0.05676 | 0.3486 15 | 15 | | -0.16 0.8728 | | 0.1 -0.6678 0.5543 | 0.5543 |

| | | | Least S | gdna | Least Squares Means | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Act<br>Tre<br>Effect (N) | Actual<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | | Lower Upper |
| GRP | 1 | 7.0175 | 0.2465 15 | 15 | 28.47 | | 0.05 | <.0001 0.05 6.4922 7.5429 | 7.5429 |
| GRP | 2 | 7.0222 | 0.2465 15 | 15 | 28.49 | | 0.05 | <.0001 0.05 6.4969 7.5476 | 7.5476 |
| GRP | 3 | 6.9608 | 0.2465 15 | 15 | 28.24 | | 0.05 | <.0001 0.05 6.4354 7.4861 | 7.4861 |

Supporting Document for Tables 15.4.3.1.1/2, 15.4.3.6.1/2, and 15.4.3.7.1/2

The Mixed Procedure

ANAL=Primary Model ANALYTEN=2 ANALYTE=Metabolite 2571107A PARM=AUC0-inf (ng\*h/mL) PARAMCD=AUCIFP

| Model Information | n |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| el<br>on | Values | 1 2 3 |
|----------------------------|--------|-------|
| Class Level<br>Information | Levels | 3 |
| D H | Class | GRP |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | Τ |
| Columns in X | 4 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 18 |

| Number of Observations | |
|-----------------------------|----|
| Number of Observations Read | 18 |
| Number of Observations Used | 18 |

| Covar<br>Paran<br>Estin | Covariance<br>Parameter<br>Estimates |
|-------------------------|--------------------------------------|
| Cov Parm | Estimate |
| Residual | 0.3549 |

| | 32.4 | 34.4 | 34.7 | 35.1 |
|---|---|---|---|---|
| Fit Statistics | -2 Res Log Likelihood | AIC (Smaller is Better) | AICC (Smaller is Better) | BIC (Smaller is Better) |

| | | Š | Solution for Fixed Effects | r Fi | xed Effe | cts | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Actual<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Intercept | | 6.9878 | 0.2432 15 | 15 | 28.73 | | 0.05 | <.0001 0.05 6.4694 7.5062 | 7.5062 |
| GRP | 1 | 0.03890 | 0.03890 0.3440 15 | 15 | | 0.11 0.9115 0.05 -0.6942 0.7720 | 0.05 | -0.6942 | 0.7720 |
| GRP | 2 | 0.04692 | 0.04692 0.3440 15 | 15 | | 0.14 0.8933 0.05 -0.6862 0.7801 | 0.05 | -0.6862 | 0.7801 |
| GRP | 3 | 0 | | | | | | | |

| iffects | Pr > F | 0.9894 |
|---------|-----------|--------|
| Fixed E | F Value | 0.01 |
| ts of | Den<br>DF | 15 |
| Tests | Num<br>DF | 2 |
| Type 3 | Effect | GRP |

| | | Est | Estimates | tes | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Standard | DF | t Value | $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | Alpha | Lower | Upper |
| Mild vs Healthy | 0.008022 | 0.008022 0.3440 15 | 15 | | 0.02 0.9817 | | 0.1 -0.5950 0.6110 | 0.6110 |
| Moderate vs Healthy -0.03890 | -0.03890 | 0.3440 15 | 15 | -0.11 | -0.11 0.9115 | 0.1 | 0.1 -0.6419 0.5641 | 0.5641 |

| | | | Least S | gana | Least Squares Means | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Actual<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha Lower Upper | Alpha | Lower | Upper |
| | 1 | 7.0267 | 0.2432 15 | 15 | 28.89 | <.0001 | 0.05 | <.0001 0.05 6.5083 7.5452 | 7.5452 |
| | 2 | 7.0348 | 0.2432 15 | 15 | 28.92 | <.0001 | 0.05 | <.0001 0.05 6.5164 7.5532 | 7.5532 |
| | 3 | 6.9878 | 0.2432 15 | 15 | 28.73 | <.0001 | 0.05 | <.0001 0.05 6.4694 7.5062 | 7.5062 |

Supporting Document for Tables 15.4.3.1.1/2, 15.4.3.6.1/2, and 15.4.3.7.1/2

The Mixed Procedure

ANAL=Primary Model ANALYTEN=2 ANALYTE=Metabolite 2571107A PARM=Cmax (ng/mL) PARAMCD=CMAX

| Model Information | no |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| el | Values | 123 |
|----------------------------|--------|-----|
| Class Level<br>Information | Levels | 3 |
| ט ב | Class | GRP |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | 1 |
| Columns in X | 4 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 18 |

| Number of Observations | |
|-----------------------------|----|
| Number of Observations Read | 18 |
| Number of Observations Used | 18 |

| | 1 | | | | | |
|--------|----|--------------|--------|-----|------|---|
| Number | οĘ | Observations | ations | Not | Used | 0 |

| Covariance Parameter Estimates Parm Estimate | 1 |
|----------------------------------------------|---|
| Covar<br>Paran<br>Estin<br>Cov Parm | 1 |

| | .3 | .3 | 9. | 0. | l |
|---|---|---|---|---|---|
| | 21.3 | 23.3 | 23.6 | 24.0 | |
| Fit Statistics | -2 Res Log Likelihood | AIC (Smaller is Better) | AICC (Smaller is Better) | BIC (Smaller is Better) | |

| | | Š | Solution for Fixed Effects | r Fi | xed Effe | cts | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Actual<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Intercept | | 2.3136 | 0.1679 15 | 15 | 13.78 | | 0.05 | <.0001 0.05 1.9557 2.6715 | 2.6715 |
| GRP | 1 | 0.3205 | 0.2374 15 | 15 | 1.35 | 1.35 0.1970 0.05 -0.1856 0.8266 | 0.05 | -0.1856 | 0.8266 |
| GRP | 2 | 0.3836 | 0.3836 0.2374 15 | 15 | 1.62 | 1.62 0.1270 0.05 -0.1225 0.8897 | 0.05 | -0.1225 | 0.8897 |
| GRP | 3 | 0 | | | | | | | |

| | | ES | Estimates | ıtes | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Standard | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Mild vs Healthy | 0.06307 | 0.2374 15 | 15 | | 0.27 0.7942 0.1 -0.3532 0.4793 | 0.1 | -0.3532 | 0.4793 |
| Moderate vs Healthy | -0.3205 | 0.2374 | 15 | -1.35 | 0.2374 15 -1.35 0.1970 0.1 -0.7368 0.09571 | 0.1 | -0.7368 | 0.09571 |

| | | | Least 5 | 3qua. | Least Squares Means | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Actual<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | $rac{1}{2} = \left \begin{array}{c c} 1 & 1 & 1 \\ \hline 1 & 1 & 1 \end{array} \right $ $\left \begin{array}{c c} 1 & 1 & 1 \\ \hline 1 & 1 & 1 \end{array} \right $ $\left \begin{array}{c c} 1 & 1 & 1 \\ \hline 1 & 1 & 1 \end{array} \right $ $\left \begin{array}{c c} 1 & 1 & 1 \\ \hline 1 & 1 & 1 \end{array} \right $ $\left \begin{array}{c c} 1 & 1 & 1 \\ \hline 1 & 1 & 1 \end{array} \right $ | Alpha | Lower | Upper |
| GRP | 1 | 2.6341 | 2.6341 0.1679 15 15.69 | 15 | 15.69 | | 0.05 | <.0001 0.05 2.2763 2.9920 | 2.9920 |
| GRP | 2 | 2.6972 | | 15 | 0.1679 15 16.07 | | 0.05 | <.0001 0.05 2.3393 3.0551 | 3.0551 |
| GRP | 3 | 2.3136 | 0.1679 15 | 15 | 13.78 | <.0001 | 0.05 | <.0001 0.05 1.9557 2.6715 | 2.6715 |

44/88

Supporting Document for Tables 15.4.3.1.1/2, 15.4.3.6.1/2, and 15.4.3.7.1/2

The Mixed Procedure

ANAL=Primary Model ANALYTEN=3 ANALYTE=Metabolite 2571109A PARM=AUCO-t (ng\*h/mL) PARAMCD=AUCLST

| Model Information | no |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| on | Values | 1 2 3 |
|----------------------------|--------|-------|
| Class Level<br>Information | Levels | 3 |
| ט ה | Class | GRP |

| 1 |
|----|
| 4 |
| 0 |
| 1 |
| 18 |

| Covariance<br>Parameter<br>Estimates | Estimate | 0.3431 |
|--------------------------------------|----------|----------|
| Covar<br>Parar<br>Estir | Cov Parm | Residual |

| Statistics | ihood 31.9 | Better) 33.9 | Better) 34.2 | Better) 34.6 |
|---|---|---|---|---|
| Fit Stat | -2 Res Log Likelihood | AIC (Smaller is E | AICC (Smaller is | BIC (Smaller is E |

| | neddn | 9.2965 10.3159 | 0.4090 | 0.2181 | |
|---|---|---|---|---|---|
| | Lower | 9.2965 | -1.0327 | -1.2236 | |
| | Alpha | 0.05 | 0.05 | 0.05 | |
| cts | ndard<br>Error DF t Value Pr > t Alpha | <.0001 0.05 | -0.92 0.3711 0.05 -1.0327 0.4090 | -1.49 0.1578 0.05 -1.2236 0.2181 | |
| ixed Effe | t Value | 41.01 | | | |
| Or<br>F | ÐΕ | 15 | 15 | 15 | |
| Solution for Fixed Effects | Standard<br>Error | 0.2391 15 | -0.3118 0.3382 15 | 0.3382 15 | |
| σ | Estimate | 9.8062 | -0.3118 | -0.5028 | 0 |
| | Actual<br>Treatment (N) | | 1 | 2 | 3 |
| | Effect | Intercept | GRP | GRP | GRP |

| ffects | Pr > F | 0.3501 |
|---------|-----------|--------|
| Fixed E | F Value | 1.13 |
| ts of | Den<br>DF | 15 |
| Test | Num<br>DF | 2 |
| Type 3 | Effect | GRP |

| | | ES1 | Estimates | tes | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Standard<br>Error | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | . Upper |
| Mild vs Healthy | -0.1909 | 0.3382 15 | 15 | -0.56 | 0.5807 | | 0.1 -0.7838 0.4019 | 0.4019 |
| Moderate vs Healthy | 0.3118 | 0.3382 15 | 15 | 0.92 | 0.3711 | | 0.1 -0.2810 0.9047 | 0.9047 |

| | | | Least | Sque | Least Squares Means | 70 | | | |
|---|---|---|---|---|---|---|---|---|---|
| Act<br>Tre<br>Effect (N) | Actual<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | Alpha | Lower | Upper |
| GRP | 1 | 9.4944 | 9.4944 0.2391 15 | 15 | 39.70 | | 0.05 | 8.9847 | <.0001 0.05 8.9847 10.0041 |
| GRP | 2 | 9.3034 | 9.3034 0.2391 15 | 15 | 38.91 | | 0.05 | 8.7937 | <.0001 0.05 8.7937 9.8131 |
| GRP | 3 | 9.8062 | 9.8062 0.2391 15 41.01 | 15 | 41.01 | | 0.05 | 9.2965 | <.0001 0.05 9.2965 10.3159 |

Supporting Document for Tables 15.4.3.1.1/2, 15.4.3.6.1/2, and 15.4.3.7.1/2

The Mixed Procedure

ANAL=Primary Model ANALYTEN=3 ANALYTE=Metabolite 2571109A PARM=AUC0-inf (ng\*h/mL) PARAMCD=AUCIFP

| Model Information | n |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| on | Values | 1 2 3 |
|----------------------------|--------|-------|
| Class Level<br>Information | Levels | 3 |
| บี่ | Class | GRP |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | 1 |
| Columns in X | 4 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 18 |

| | Z | Number of Observations | |
|----------|----|------------------------|----|
| Number o | of | Observations Read | 18 |
| Number o | of | Observations Used | 18 |

| | O | 0 |
|--------------------------------------|----------|----------|
| covariance<br>Parameter<br>Estimates | Estimate | 0.3420 |
| Covar<br>Parar<br>Estir | Cov Parm | Residual |

| Statistics | lhood 31.8 | is Better) 33.8 | Better) 34.2 | Better) 34.6 |
|---|---|---|---|---|
| Fit Stati | -2 Res Log Likelihood | AIC (Smaller is Be | AICC (Smaller is ] | BIC (Smaller is Be |

| | | Ø | Solution for Fixed Effects | or F: | ixed Effe | cts | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Actual<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Intercept | | 9.8232 | 0.2387 15 | 15 | 41.15 | | 90.0 | <.0001 0.05 9.3143 10.3320 | 10.3320 |
| GRP | 1 | -0.3185 | 0.3376 15 | 15 | | -0.94 0.3604 0.05 -1.0382 0.4011 | 90.0 | -1.0382 | 0.4011 |
| GRP | 2 | -0.5127 | 0.3376 15 | 15 | -1.52 | 0.1497 0.05 -1.2323 | 90.0 | -1.2323 | 0.2069 |
| GRP | 3 | 0 | | | | | | | |

| fects | Pr > F | 0.3355 |
|----------|-----------|--------|
| Fixed Ef | F Value | 1.18 |
| cs of | Den<br>DF | 15 |
| Test | Num<br>DF | 2 |
| Type 3 | Effect | GRP |

| | | Est | Estimates | tes | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Standard | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Mild vs Healthy | -0.1942 | 0.3376 15 | 15 | -0.58 | 0.5738 | 0.1 | 0.1 -0.7860 0.3977 | 0.3977 |
| Moderate vs Healthy | 0.3185 | 0.3376 15 | 15 | 0.94 | 0.3604 | | 0.1 -0.2733 0.9104 | 0.9104 |

| | | | Least | Sque | Least Squares Means | τΩ | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Actual<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | Alpha | Lower | Upper |
| GRP | 1 | 9.5046 | 9.5046 0.2387 15 | 15 | 39.81 | | 0.05 | 8.9958 | <.0001 0.05 8.9958 10.0135 |
| GRP | 2 | 9.3105 | 0.2387 15 | 15 | 39.00 | | 90.0 | 8.8016 | <.0001 0.05 8.8016 9.8193 |
| GRP | 3 | 9.8232 | 0.2387 15 | 15 | 41.15 | | 90.0 | 9.3143 | <.0001 0.05 9.3143 10.3320 |

Supporting Document for Tables 15.4.3.1.1/2, 15.4.3.6.1/2, and 15.4.3.7.1/2

The Mixed Procedure

ANAL=Primary Model ANALYTEN=3 ANALYTE=Metabolite 2571109A PARM=Cmax (ng/mL) PARAMCD=CMAX

| Model Information | n |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| el<br>on | Values | 1 2 3 |
|----------------------------|--------|-------|
| Class Level<br>Information | Levels | 3 |
| υĤ | Class | GRP |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | 1 |
| Columns in X | 4 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 18 |

| Number of Observations | |
|-----------------------------|----|
| Number of Observations Read | 18 |
| Number of Observations Used | 18 |

| Covariance<br>Parameter | Estimates | Estimate | 0.1481 |
|-------------------------|-----------|----------|----------|
| Covar | Estir | Cov Parm | Residual |

| -2 Res Log Likelihood 19.3 AIC (Smaller is Better) 21.3 AICC (Smaller is Better) 21.6 BIC (Smaller is Better) 22.0 | Fit Statistics | |
|---|---|---|
| is Better) r is Better) is Better) | es Log Likelihood | 19.3 |
| (Smaller is Better) | | 21.3 |
| is Better) | | 21.6 |
| | 1.8 | 22.0 |

| | | Š | Solution for Fixed Effects | r<br>Fi | xed Effe | cts | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Actual<br>Treatment (N) | Estimate | Standard<br>Error | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | | Lower Upper |
| Intercept | | 5.1042 | 0.1571 15 | 15 | 32.49 | <.0001 | 0.05 | <.0001 0.05 4.7693 5.4391 | 5.4391 |
| GRP | 1 | -0.1380 | -0.1380 0.2222 15 -0.62 0.5438 0.05 -0.6116 0.3356 | 15 | -0.62 | 0.5438 | 0.05 | -0.6116 | 0.3356 |
| GRP | 2 | -0.2181 | -0.2181 0.2222 15 -0.98 0.3418 0.05 -0.6918 0.2555 | 15 | -0.98 | 0.3418 | 0.05 | -0.6918 | 0.2555 |
| GRP | 3 | 0 | | | | | | | |

| ffects | Pr > F | 0.6202 |
|----------|-----------|--------|
| Fixed Ef | F Value | 0.49 |
| cs of | Den<br>DF | 15 |
| Tests | Num<br>DF | 2 |
| Type 3 | Effect | GRP |

| | | Est | Estimates | tes | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Standard | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Mild vs Healthy | -0.08011 | 0.2222 15 | 15 | -0.36 | 0.7235 | | 0.1 -0.4696 0.3094 | 0.3094 |
| Moderate vs Healthy | 0.1380 | 0.2222 15 | 15 | 0.62 | 0.5438 | | 0.1 -0.2515 0.5276 | 0.5276 |

| | | | Least S | iqua | Least Squares Means | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Act<br>Tre<br>Effect (N) | Actual<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | $\frac{1}{2}$ and $\frac{1}{2}$ | Alpha | Lower | reddn |
| GRP | 1 | 4.9662 | | 15 | 31.61 | 0.1571 15 31.61 <.0001 0.05 4.6313 5.3011 | 0.05 | 4.6313 | 5.3011 |
| GRP | 2 | 4.8861 | | 15 | 0.1571 15 31.10 | <.0001 0.05 4.5512 5.2210 | 0.05 | 4.5512 | 5.2210 |
| GRP | 3 | 5.1042 | 0.1571 | 15 | 0.1571 15 32.49 | | 0.05 | <.0001 0.05 4.7693 5.4391 | 5.4391 |

Supporting Document for Tables 15.4.3.2.1/2

The Mixed Procedure

ANAL=Additional Model 1 ANALYTEN=1 ANALYTE=Tepotinib PARM=AUCO-t (ng\*h/mL) PARAMCD=AUCLST

| Model Information | n |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| el<br>on | Values | 1 2 3 | F M |
|----------------------------|--------|-------|-----|
| Class Level<br>Information | Levels | 3 | 2 |
| D H | Class | GRP | XEX |

| | 1 | 8 | 0 | 1 | 18 |
|---|---|---|---|---|---|
| Dimensions | Covariance Parameters | Columns in X | Columns in Z | Subjects | Max Obs per Subject |

| | 18 |
|------------------------|-----------------------------|
| Number of Observations | Number of Observations Read |

| ter | Estimate | 0.1353 |
|------------------------|----------|----------|
| Parameter<br>Estimates | Cov Parm | Residual |

| | 31.2 | 33.2 | 33.6 | 33.7 |
|---|---|---|---|---|
| Fit Statistics | -2 Res Log Likelihood | AIC (Smaller is Better) | AICC (Smaller is Better) | BIC (Smaller is Better) |

| | | | Sol | Solution for Fixed Effects | Fix | ed Effect | ŭ | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | Actual<br>Treatment<br>(N) | Estimate | Standard | DF | t Value | Pr > t | Alpha | Lower | Upper |
| Intercept | | | 8069.8 | 0.8762 | 12 | 9.92 | <.0001 | 0.05 | 6.7816 | 10.6000 |
| GRP | | 1 | 0.1863 | 0.2154 | 12 | 0.87 | 0.4039 | 0.05 | -0.2829 | 9559.0 |
| GRP | | 2 | 0.001881 | 0.2223 | 12 | 0.01 | 0.9934 | 0.05 | -0.4824 | 0.4862 |
| GRP | | 3 | 0 | | | | | | | |
| SEX | Ē | | 0.2845 | 0.2210 | 12 | 1.29 | 0.2224 | 0.05 | 1791.0- | 0992.0 |
| SEX | M | | 0 | | | | | | | |
| AGE | | | 0.02540 | 0.01327 | 12 | 1.91 | 0.0797 | 0.05 | -0.00351 | 0.05431 |
| BLWEIGHT | | | -0.00224 | 0.007054 | 12 | -0.32 | 0.7567 | 0.05 | -0.01761 0.01313 | 0.01313 |

| fects | 4 < 14 | 0.6442 | 0.2224 | 0.0797 | 0.7567 |
|------------------|-----------|--------|--------|--------|----------|
| of Fixed Effects | F Value | 0.46 | 1.66 | 29.8 | 01.0 |
| o E | Den | 12 | 12 | 12 | 12 |
| Tests | Num<br>DF | 2 | Τ | 1 | Τ |
| Type 3 | Effect | GRP | XIS | AGE | BLWEIGHT |

| | | EST | - IIII | Estimates | | | | |
|---|---|---|---|---|---|---|---|---|
| Est | Estimate | Standard<br>Error | DF | t Value | ndard Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Mild vs Healthy -0 | -0.1845 | 0.2333 12 | 12 | | -0.79 0.4445 0.1 -0.6003 0.2314 | 0.1 | -0.6003 | 0.2314 |
| Moderate vs Healthy -0 | -0.1863 | 0.2154 12 | 12 | | -0.87 0.4039 0.1 -0.5702 0.1975 | 0.1 | -0.5702 | 0.1975 |

| | | | Least | Sque | Least Squares Means | D | | | |
|---|---|---|---|---|---|---|---|---|---|
| Act<br>Tre<br>Effect (N) | Actual<br>Treatment<br>(N) | Estimate | Sta | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha Lower | Alpha | Lower | Upper |
| GRP | 1 | 10.3427 | 10.3427 0.1718 12 | 12 | 60.21 | | 0.05 | 9.9684 | <.0001 0.05 9.9684 10.7169 |
| GRP | 2 | 10.1582 | 10.1582 0.1634 12 62.17 | 12 | 62.17 | | 0.05 | 9.8022 | <.0001 0.05 9.8022 10.5142 |
| GRP | 3 | 10.1563 | 10.1563 0.1666 12 60.98 | 12 | 60.98 | | 0.05 | 9.7934 | <.0001 0.05 9.7934 10.5192 |

Supporting Document for Tables 15.4.3.2.1/2

The Mixed Procedure

ANAL=Additional Model 1 ANALYTEN=1 ANALYTE=Tepotinib PARM=AUC0-inf (ng\*h/mL) PARAMCD=AUCIFP

| Model Information | no |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| el<br>on | Values | 1 2 3 | 2 F M |
|----------------------------|--------|-------|-------|
| Class Level<br>Information | Levels | 3 | 2 |
| D H | Class | GRP | SEX |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | 1 |
| Columns in X | 8 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 18 |

| | 18 |
|------------------------|-----------------------------|
| Number of Observations | Number of Observations Read |

| | 18 | 0 |
|---|---|---|
| Number of Observations | Number of Observations Used | Number of Observations Not Used |

| | 4) | |
|--------------------------------------|----------|----------|
| Covarlance<br>Parameter<br>Estimates | Estimate | 0.1290 |
| Covar<br>Parar<br>Estir | Cov Parm | Residual |

| | 30.6 | 32.6 | 33.0 | 33.1 |
|---|---|---|---|---|
| Fit Statistics | -2 Res Log Likelihood | AIC (Smaller is Better) | AICC (Smaller is Better) | BIC (Smaller is Better) |

| | | | Sol | Solution for Fixed Effects | Fix | ed Effect | Ø | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | Actual<br>Treatment<br>(N) | Estimate | Standard | DF | | t Value Pr > t | Alpha | Lower | Upper |
| Intercept | | | 8.7302 | 0.8555 | 12 | 10.21 | <.0001 | 0.05 | 6.8663 | 10.5941 |
| GRP | | 1 | 0.1766 | 0.2103 | 12 | 0.84 | 0.4173 | 0.05 | -0.2815 | 0.6348 |
| GRP | | 2 | -0.00247 | 0.2170 | 12 | -0.01 | 1166.0 | 0.05 | -0.4753 | 0.4704 |
| GRP | | 3 | 0 | | | | | | | |
| SEX | 댼 | | 0.2832 | 0.2158 | 12 | 1.31 | 0.2140 | 0.05 | -0.1870 | 0.7533 |
| SEX | М | | 0 | | | | | | | |
| AGE | | | 0.02489 | 0.01295 | 12 | 1.92 | 0.0787 | 0.05 | -0.00333 0.05312 | 0.05312 |
| BLWEIGHT | | | -0.00205 | 0.006887 | 12 | -0.30 | 0.7714 | 0.05 | -0.01705 0.01296 | 0.01296 |

| TESTS OF FIXER BLIECTS |
|------------------------|
| Den<br>DF |
| 12 |
| 12 |
| 12 |
| 12 |

| | | ES1 | Estimates | tes | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Standard<br>Error | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Mild vs Healthy | -0.1791 | | 12 | -0.79 | 0.2278 12 -0.79 0.4470 0.1 -0.5851 0.2269 | 0.1 | -0.5851 | 0.2269 |
| Moderate vs Healthy | -0.1766 | -0.1766 0.2103 12 -0.84 0.4173 0.1 -0.5514 0.1981 | 12 | -0.84 | 0.4173 | 0.1 | -0.5514 | 0.1981 |

| | | | Least | Sque | Least Squares Means | ω | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Actual<br>Treatment<br>(N) | Estimate | Sta | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha Lower | Alpha | Lower | Upper |
| GRP | 1 | 10.3580 | 10.3580 0.1677 12 61.77 | 12 | 61.77 | | 0.05 | 9.9926 | <.0001 0.05 9.9926 10.7234 |
| GRP | 2 | 10.1789 | 0.1595 | 12 | 0.1595 12 63.81 | | 0.05 | 9.8313 | <.0001 0.05 9.8313 10.5265 |
| GRP | 3 | 10.1814 | 10.1814 0.1626 12 62.61 | 12 | 62.61 | l | 0.05 | 9.8271 | <.0001 0.05 9.8271 10.5357 |

Supporting Document for Tables 15.4.3.2.1/2

The Mixed Procedure

ANAL=Additional Model 1 ANALYTEN=1 ANALYTE=Tepotinib PARM=Cmax (ng/mL) PARAMCD=CMAX

| Model Information | n |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| el<br>on | Values | 123 | F M |
|----------------------------|--------|-----|-----|
| Class Level<br>Information | Levels | 3 | 2 |
| БЦ | Class | GRP | SEX |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | 1 |
| Columns in X | 8 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 18 |

| | 18 |
|------------------------|-----------------------------|
| Number of Observations | Number of Observations Read |

| Number of Observations | |
|---------------------------------|----|
| Number of Observations Used | 18 |
| Number of Observations Not Used | 0 |

| Covariance<br>Parameter<br>Estimates | Estimate | 0.05446 |
|--------------------------------------|----------|----------|
| Covai<br>Parar<br>Estir | Cov Parm | Residual |

| | 20.3 | 22.3 | 7.22 | 22.7 |
|---|---|---|---|---|
| Fit Statistics | -2 Res Log Likelihood | AIC (Smaller is Better) | AICC (Smaller is Better) | BIC (Smaller is Better) |

| | | | So | Solution for Fixed Effects | Fix | red Effec | ts | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | Actual<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Tower | Upper |
| Intercept | | | 4.9944 | 0.5558 | 12 | 8.99 | <.0001 | 0.05 | 3.7833 | 6.2055 |
| GRP | | 1 | 0.3604 | 0.1366 | 12 | 2.64 | 0.0217 | 0.05 | 0.06269 | 0.6581 |
| GRP | | 7 | 0.3267 | 0.1410 | 12 | 2.32 | 0.0390 | 0.05 | 0.01950 | 0.6339 |
| GRP | | 3 | 0 | | | | | | | |
| SEX | 伍 | | 0.1918 | 0.1402 | 12 | 1.37 | 0.1964 | 0.05 | -0.1137 | 0.4973 |
| SEX | М | | 0 | | | | | | | |
| AGE | | | 0.01072 | 0.008416 | 12 | 1.27 | 0.2270 | 0.05 | -0.00762 | 0.02905 |
| BLWEIGHT | | | 80000.0- | 0.004475 | 12 | -0.02 | 0.9863 | 0.05 | .00083 | 0.009671 |

| fects | Fr > F | 0.0384 | 0.1964 | 0.2270 | 0.00 |
|------------------|-----------|--------|--------|--------|----------|
| of Fixed Effects | F Value | 4.33 | 1.87 | 1.62 | 00.0 |
| s of | Den | 12 | 12 | 12 | 12 |
| Test | Num<br>DF | 2 | 1 | 1 | 1 |
| Type 3 Tests | Effect | GRP | SEX | AGE | BLWEIGHT |

| | | EB | Estimates | ıtes | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Standard | DF | t Value | ndard Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Mild vs Healthy | -0.03366 | -0.03366 0.1480 12 | 12 | | -0.23 0.8239 0.1 -0.2974 0.2301 | 0.1 | -0.2974 | 0.2301 |
| Moderate vs Healthy | -0.3604 | -0.3604 0.1366 12 -2.64 0.0217 0.1 -0.6039 -0.1169 | 12 | -2.64 | 0.0217 | 0.1 | -0.6039 | -0.1169 |

| | ләбб | 6.3224 | 6.2772 | 5.9548 |
|---|---|---|---|---|
| | Lower | <.0001 0.05 5.8476 6.3224 | <.0001 0.05 5.8255 6.2772 | <.0001 0.05 5.4944 5.9548 |
| | Alpha | 90.0 | 90.0 | 0.05 |
| | ndard<br>Error DF t Value Pr > t Alpha | <.0001 | <.0001 | <.0001 |
| Least Squares Means | t Value | 55.85 | 58.38 | 54.18 |
| igua | DF | 12 | 12 | 12 |
| Least 8 | Standard<br>Error | 0.1090 12 | 6.0514 0.1036 12 | 5.7246 0.1057 12 54.18 |
| | Estimate | 6.0850 | 6.0514 | 5.7246 |
| | Actual<br>Treatment<br>(N) | 1 | 2 | 3 |
| | Effect | GRP | GRP | GRP |

Supporting Document for Tables 15.4.3.3.1/2

The Mixed Procedure

ANAL=Additional Model 2 ANALYTEN=1 ANALYTE=Tepotinib PARM=AUCO-t (ng\*h/mL) PARAMCD=AUCLST

| Model Information | no |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| rel | Values | 1 2 | F M |
|----------------------------|--------|-----|-----|
| Class Level<br>Information | Levels | 2 | 2 |
| D H | Class | GRP | SEX |

| | 1 | 7 | 0 | 1 | 18 |
|---|---|---|---|---|---|
| Dimensions | Covariance Parameters | Columns in X | Columns in Z | Subjects | Max Obs per Subject |

| Number of Observations | |
|----------------------------|----|
| umber of Observations Read | 18 |

| | Z | Number of Observations | bservation | ĽΩ | |
|----------|----|---------------------------------|------------|----|----|
| Number c | υĘ | Number of Observations Used | ns Used | | 18 |
| Number c | ΣĘ | Number of Observations Not Used | ns Not Use | pa | 0 |
| | | Covariance<br>Parameter | iance | | |
| | | Estimates | lates | | |
| | | Cov Parm | Estimate | | |
| | | Residual | 0.1329 | | |

| Parameter<br>Estimates | rm Estimate | al 0.1329 |
|------------------------|-------------|-----------|
| Parame<br>Estima | Cov Parm | Residual |

| | 30.7 | 32.7 | 33.1 | 33.3 |
|---|---|---|---|---|
| Fit Statistics | -2 Res Log Likelihood | AIC (Smaller is Better) | AICC (Smaller is Better) | BIC (Smaller is Better) |

| | | | | Solution for Fixed Effects | for | Fixed Ef | fects | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | GRP | Estimate | Standard<br>Error DF | DF | t Value | t Value $ Pr > t $ Alpha | Alpha | Lower | ләddn |
| Intercept | | | 8.7925 | 0.8576 13 | 13 | 10.25 | <.0001 | 0.05 | | 6.9398 10.6452 |
| GRP | | П | 0.07693 | 0.1980 | 13 | 0.39 | 0.7040 | 0.05 | -0.3509 | 0.5048 |
| GRP | | 7 | 0 | | | | | | | |
| XES | ĒΨ | | 0.2610 | 0.2177 13 | 13 | 1.20 | 0.2519 | 0.05 | -0.2093 | 0.7313 |
| XES | М | | 0 | | | | | | | |
| AGE | | | 0.02202 | 0.01279 13 | 13 | 1.72 | | 0.05 | 0.1087 0.05 -0.00561 0.04965 | 0.04965 |
| BLWEIGHT | | | -0.00095 | -0.00095 0.006651 13 | 13 | -0.14 | 0.8883 | | 0.05 -0.01532 0.01342 | 0.01342 |
| | | | | | | | | | | ۱ |

Type 3 Tests of Fixed Effects

| Pr > F | 0.7040 | 0.2519 | 0.1087 | 0.8883 |
|-----------|--------|--------|--------|----------|
| F Value | 0.15 | 1.44 | 2.97 | 0.02 |
| Den<br>DF | 13 | 13 | 13 | 13 |
| Num<br>DF | 1 | 1 | 1 | 1 |
| Effect | GRP | SEX | AGE | BLWEIGHT |

| | | EB | tima | Estimates | | | | |
|---|---|---|---|---|---|---|---|---|
| abel | Estimate | Standard | DF | t Value | ndard Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| | | | | 3 | ' | <u>F</u> | 1 | 1 (1) |
| Grade 2 vs Grade 1 | -0.07693 | 0.1980 13 | 13 | | -0.39 0.7040 | | 0.1 -0.4276 0.2738 | 0.2738 |

| | | | Lea | ist 5 | Least Squares M | Means | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Standard | | | | | | |
| Effect | GRP | Effect GRP Estimate | Error | DF | t Value | Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| GRP | 1 | 10.2339 | 0.1155 13 | 13 | 88.57 | | 0.05 | 9.9843 | <.0001 0.05 9.9843 10.4836 |
| GRP | 2 | 10.1570 | 0.1826 13 | 13 | 55.61 | | 0.05 | 9.7624 | <.0001 0.05 9.7624 10.5516 |

Supporting Document for Tables 15.4.3.3.1/2

The Mixed Procedure

ANAL=Additional Model 2 ANALYTEN=1 ANALYTE=Tepotinib PARM=AUC0-inf (ng\*h/mL) PARAMCD=AUCIFP

| Model information | n |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| el | Values | 1 2 | ЫM |
|----------------------------|--------|-----|-----|
| Class Level<br>Information | Levels | 2 | 2 |
| | Class | GRP | SEX |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | 1 |
| Columns in X | 7 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 18 |

| Number of Observations | |
|-----------------------------|----|
| Number of Observations Read | 18 |

| | 18 | 0 |
|---|---|---|
| Number of Observations | Number of Observations Used | Number of Observations Not Used |

| ns Used | of Observations Not Used | Covariance | Parameter<br>Estimates | Estimate | 0.1264 |
|---|---|---|---|---|---|
| ot Observations | Observatic | Covar | Paran<br>Estin | Cov Parm | Residual |
| O<br>H | oĘ | | | | |

| | 30.1 | 32.1 | 32.4 | 32.6 |
|---|---|---|---|---|
| Fit Statistics | -2 Res Log Likelihood | AIC (Smaller is Better) | AICC (Smaller is Better) | BIC (Smaller is Better) |

| | | | | Solution for Fixed Effects | for | Fixed Ef: | fects | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | GRP | Estimate | Standard<br>Error DF | DF | t Value | t Value $ Pr > t Alpha$ | Alpha | Lower | ләddn |
| Intercept | | | 8.8252 | 0.8362 13 | 13 | 10.55 | | <.0001 0.05 | | 7.0186 10.6318 |
| GRP | | 1 | 0.07404 | 0.1931 13 | 13 | 0.38 | 0.7076 | 0.05 | -0.3432 | 0.4912 |
| GRP | | 7 | 0 | | | | | | | |
| XES | দ | | 0.2601 | 0.2123 | 13 | 1.23 | 0.2422 | 0.05 | -0.1985 | 0.7187 |
| XES | М | | 0 | | | | | | | |
| AGE | | | 0.02162 | 0.01247 13 | 13 | 1.73 | 0.1066 | 0.05 | 0.05 -0.00532 0.04856 | 0.04856 |
| BLWEIGHT | | | -0.00079 | -0.00079 0.006486 13 | 13 | -0.12 | | 0.05 | 0.9051 0.05 -0.01480 0.01322 | 0.01322 |

Type 3 Tests of Fixed Effects

| Effect | Num | Den<br>DF | F Value | Pr > F |
|----------|-----|-----------|---------|--------|
| GRP | 1 | 13 | 0.15 | 0.7076 |
| SEX | 1 | 13 | 1.50 | 0.2422 |
| AGE | 1 | 13 | 3.01 | 9901.0 |
| BLWEIGHT | 1 | 13 | 10.0 | 0.9051 |

| | | E<br>E | time | Estimates | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Standard | | | | | | |
| Label | Estimate | Error | DF | t Value | Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Grade 2 vs Grade 1 -0.07404 | -0.07404 | 0.1931 13 | 13 | -0.38 | -0.38 0.7076 | | 0.1 -0.4160 0.2680 | 0.2680 |

| | ч | 0 | т |
|---|---|---|---|
| | Lower Upper | 10.497 | 10.564 |
| | | <.0001 0.05 10.0102 10.4970 | <.0001 0.05 9.7948 10.5643 |
| | Alpha | 0.05 | 0.05 |
| leans | ndard<br>Error DF t Value Pr > t Alpha | | |
| Least Squares Means | t Value | 0.1127 13 91.01 | 57.16 |
| ast | DF | 13 | 13 |
| Le | Standard<br>Error | 0.1127 | 10.1796 0.1781 13 57.16 |
| | Effect GRP Estimate | 10.2536 | 10.1796 |
| | GRP | 1 | 2 |
| | Effect | GRP | GRP |

Supporting Document for Tables 15.4.3.3.1/2

The Mixed Procedure

ANAL=Additional Model 2 ANALYTEN=1 ANALYTE=Tepotinib PARM=Cmax (ng/mL) PARAMCD=CMAX

| Model Information | no |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| el | Values | 1 2 | 2 F M |
|----------------------------|--------|-----|-------|
| Class Level<br>Information | Levels | 2 | 2 |
| 13 E | Class | GRP | SEX |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | 1 |
| Columns in X | 7 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 18 |

| Number of Observations | |
|-----------------------------|----|
| Number of Observations Read | 18 |

| | 18 | 0 |
|---|---|---|
| Number of Observations | Number of Observations Used | Number of Observations Not Used |

| | - | |
|--------------------------------------|----------|----------|
| covariance<br>Parameter<br>Estimates | Estimate | 0.05782 |
| Covar<br>Parar<br>Estir | Cov Parm | Residual |

| | 19.9 | 21.9 | 22.3 | 22.5 |
|---|---|---|---|---|
| Fit Statistics | -2 Res Log Likelihood | AIC (Smaller is Better) | AICC (Smaller is Better) | BIC (Smaller is Better) |

| | | | | Solution for Fixed Effects | for | Fixed Ef | fects | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | GRP | Estimate | Standard<br>Error DF | | t Value | t Value Pr > t Alpha | Alpha | Lower | Upper |
| Intercept | | | 5.3831 | 0.5657 | 13 | 9.52 | <.0001 | 0.05 | 4.1610 | 6.6052 |
| GRP | | П | 0.3320 | 0.1306 | 13 | 2.54 | 0.0246 | 90.0 | 0.04981 | 0.6143 |
| GRP | | 7 | 0 | | | | | | | |
| SEX | ĒΉ | | 0.1793 | 0.1436 | 13 | 1.25 | 0.2338 | 90.0 | -0.1309 | 0.4896 |
| SEX | М | | 0 | | | | | | | |
| AGE | | | 0.007516 | 0.007516 0.008436 | 13 | 0.89 | 0.3892 | | 0.05 -0.01071 | 0.02574 |
| BLWEIGHT | | | -0.00241 | -0.00241 0.004387 13 | 13 | -0.55 | 0.5916 | | 0.05 -0.01189 0.007065 | 0.007065 |

Type 3 Tests of Fixed Effects

| ffect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|----------|-----------|-----------|---------|--------|
| GRP | 1 | 13 | 6.46 | 0.0246 |
| SEX | 1 | 13 | 1.56 | 0.2338 |
| AGE | 1 | 13 | 0.79 | 0.3892 |
| BLWEIGHT | 1 | 13 | 0.30 | 0.5916 |

| | | | Leas | st S | Least Squares Means | ans | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect GRP | GRP | Estimate | Standard | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | | Lower Upper |
| GRP | 1 | 6.0424 | 6.0424 0.07622 13 | 13 | 79.28 | | 0.05 | <.0001 0.05 5.8778 6.2071 | 6.2071 |
| GRP | 2 | 5.7104 | 0.1205 13 | 13 | 47.40 | 47.40 <.0001 0.05 5.4501 5.9707 | 0.05 | 5.4501 | 2.9707 |

Supporting Document for Tables 15.4.3.4.1/2

The Mixed Procedure

ANAL=Additional Model 3 ANALYTEN=1 ANALYTE=Tepotinib PARM=AUCO-t (ng\*h/mL) PARAMCD=AUCLST

| Model Information | no |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| | 70 | 4 | |
|----------------------------|--------|----------|-----|
| | 168 | 3 4 | |
| | Values | 7 | Σ |
| re]<br>[or | Va | $\vdash$ | ſΞų |
| Class Level<br>Information | Levels | 4 | 2 |
| I O | Class | GRP | SEX |

| Number of Observations | |
|----------------------------|----|
| umber of Observations Read | 18 |

| 18 | 0 |
|-----------------------------|---------------------------------|
| Number of Observations Used | Number of Observations Not Used |

| | O. | œ |
|--------------------------------------|----------|----------|
| covariance<br>Parameter<br>Estimates | Estimate | 80580.0 |
| Covar<br>Paran<br>Estin | Cov Parm | Residual |

| | 24.2 | 26.2 | 7.92 | 26.6 |
|---|---|---|---|---|
| Fit Statistics | -2 Res Log Likelihood | AIC (Smaller is Better) | AICC (Smaller is Better) | BIC (Smaller is Better) |

| Solution for Fixed Effects |
|----------------------------|
| Standard Estimate Error |
| 9.3885 0.7424 |
| -0.1884 0.3126 |
| -0.6956 0.3290 |
| -0.2941 0.3782 |
| 0 |
| 0.2710 0.1777 |
| 0 |
| 0.01568 0.01134 |
| 0.000633 0.005388 |
| _ | | | | | |
|--------------|-----------|--------|--------|--------|----------|
| | Fr > F | 0.0671 | 0.1556 | 0.1942 | 9806.0 |
| race Erreces | F Value | 3.18 | 2.32 | 1.91 | 0.01 |
| o<br>I | Den | 11 | 11 | 11 | 11 |
| 1000 | Num<br>DF | 3 | 1 | 1 | Τ |
| TABE 3 | Effect | GRP | SEX | AGE | BLWEIGHT |

| | | Ä | stim | Estimates | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Standard | DF | t Value | ndard Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Mild vs Normal | -0.5072 | -0.5072 0.1779 11 | 11 | | -2.85 0.0158 | | 0.1 -0.8266 -0.1877 | -0.1877 |
| Moderate vs Normal | -0.1057 | -0.1057 0.2401 11 | 11 | -0.44 | -0.44 0.6684 0.1 -0.5369 0.3256 | 0.1 | -0.5369 | 0.3256 |
| Severe vs Normal | 0.1884 | 0.1884 0.3126 11 | 11 | | 0.60 0.5588 | | 0.1 -0.3729 0.7498 | 0.7498 |

| | | | Lea | ast | Least Squares Means | <b>l</b> eans | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | GRP | Effect GRP Estimate | Standard | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | |
| GRP | 1 | 10.3293 | 10.3293 0.09690 11 106.59 | 11 | 106.59 | | 0.05 | <.0001 0.05 10.1160 10.5426 | 10.5426 |
| GRP | 2 | 9.8222 | | 11 | 0.1600 11 61.39 | | 0.05 | <.0001 0.05 9.4700 10.1743 | 10.1743 |
| GRP | 3 | 10.2237 | 10.2237 0.2364 11 43.24 | 11 | 43.24 | | 0.05 | <.0001 0.05 9.7032 10.7441 | 10.7441 |
| GRP | 4 | 10.5177 | 10.5177 0.3078 11 34.17 | 11 | 34.17 | | 0.05 | <.0001 0.05 9.8402 11.1953 | 11.1953 |

Supporting Document for Tables 15.4.3.4.1/2

The Mixed Procedure

ANAL=Additional Model 3 ANALYTEN=1 ANALYTE=Tepotinib PARM=AUC0-inf (ng\*h/mL) PARAMCD=AUCIFP

| Model Information | no |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| | 70 | 4 | |
|----------------------------|--------|------|-----|
| | Values | 1234 | |
| | alı | 0 | Σ |
| re] | 5 | Н | F M |
| Class Level<br>Information | Levels | 4 | 2 |
| ОН | Class | GRP | SEX |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | Τ |
| Columns in X | 6 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 18 |

| Number of Observations | |
|-----------------------------|----|
| Number of Observations Read | 18 |

75/88

| Number of Observations Number of Observations Used Number of Observations Not Used 0 | | | |
|---|---|---|---|
| Number of Observat: of Observations Used of Observations Not | | 18 | 0 |
| | Observation | of Observations | of Observations Not |

| Covariance<br>Parameter<br>Estimates | Estimate | 0.08325 |
|--------------------------------------|----------|----------|
| Covarianc<br>Paramete<br>Estimate | Cov Parm | Residual |

| | 24.0 | 26.0 | 26.4 | 26.4 |
|---|---|---|---|---|
| Fit Statistics | -2 Res Log Likelihood | AIC (Smaller is Better) | AICC (Smaller is Better) | BIC (Smaller is Better) |

| 3 | 51 | 01 | Solution for Fixed Effects | for | Fixed Ef | fects | | | |
|---|---|---|---|---|---|---|---|---|---|
| Sex GRP Estimate Error | Sta<br>Estimate | Standar<br>Erro | ъ́й | DF | t Value | Pr > t | Alpha | Lower | Upper |
| 9.3997 0.7343 | | 0.734 | 33 | 11 | 12.80 | <.0001 | 90.0 | 7.7835 | 11.0159 |
| 1 -0.1909 0.3092 | | 30ε·0 | 92 | 11 | -0.62 | 0.5495 | 0.05 | -0.8713 | 0.4896 |
| 2 -0.6743 0.3254 | | 0.32 | 54 | 11 | -2.07 | 0.0625 | 90.0 | -1.3905 | 0.04188 |
| 3 -0.2966 0.3741 | | LE.0 | 41 | 11 | 62.0- | 0.4447 | 90.0 | -1.1201 | 0.5269 |
| 4 0 | 0 | | | | | | | | |
| F 0.2699 0.1758 | | 0.17 | 58 | 11 | 1.54 | 0.1530 | 90.0 | -0.1170 | 0.6569 |
| 0 M | 0 | | | | | | | | |
| 0.01571 0.01122 | | 0.01 | 122 | 11 | 1.40 | 0.1890 | 0.05 | -0.00898 | 0.04040 |
| 0.000689 0.005330 | | | 330 | 11 | 0.13 | 0.8994 | 0.05 | -0.01104 | 0.01242 |

| 1 YPG 0 | בת<br>ה<br>ה | 5 | FINGS EL | EL LACCES |
|----------|--------------|-----|----------|-----------|
| Effect | Num<br>DF | Den | F Value | Pr > F |
| GRP | 3 | 11 | 2.99 | 0.0777 |
| SEX | 1 | 11 | 2.36 | 0.1530 |
| AGE | 1 | 11 | 1.96 | 0.1890 |
| BLWEIGHT | 1 | 11 | 0.02 | 0.8994 |

| | | Ä | stim | Estimates | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Standard | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Mild vs Normal | -0.4834 | -0.4834 0.1759 11 | 11 | | -2.75 0.0190 0.1 -0.7994 -0.1675 | 0.1 | -0.7994 | -0.1675 |
| Moderate vs Normal | -0.1057 | 0.2375 | 11 | -0.45 | -0.1057 0.2375 11 -0.45 0.6648 0.1 -0.5323 0.3208 | 0.1 | -0.5323 | 0.3208 |
| Severe vs Normal | 0.1909 | 0.1909 0.3092 11 | 11 | | 0.62 0.5495 | 0.1 | 0.1 -0.3643 0.7461 | 0.7461 |

| | | | Lea | ast | Least Squares Means | leans | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect GRP | GRP | Estimate | Standard | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | томег | $_{ m A}$ |
| GRP | 1 | 10.3443 | 10.3443 0.09585 11 107.92 | 11 | 107.92 | <.0001 | 0.05 | <.0001 0.05 10.1334 10.5553 | 10.5553 |
| GRP | 7 | 6098.6 | 0.1583 11 | 11 | 62.31 | <.0001 | 0.05 | <.0001 0.05 9.5125 10.2092 | 10.2092 |
| GRP | 3 | 10.2386 | | 11 | 0.2339 11 43.78 | <.0001 | 0.05 | <.0001 0.05 9.7238 10.7534 | 10.7534 |
| GRP | 4 | 10.5352 | | 11 | 0.3045 11 34.60 | | 0.05 | <.0001 0.05 9.8650 11.2054 | 11.2054 |

Supporting Document for Tables 15.4.3.4.1/2

The Mixed Procedure

ANAL=Additional Model 3 ANALYTEN=1 ANALYTE=Tepotinib PARM=Cmax (ng/mL) PARAMCD=CMAX

| Model Information | n |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| | 70 | 4 | |
|----------------------------|--------|----------|-----|
| | 168 | m | |
| | Values | 1234 | Σ |
| re] | 5 | $\vdash$ | F M |
| Class Level<br>Information | Levels | 4 | 2 |
| ОП | Class | GRP | SEX |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | 1 |
| Columns in X | 6 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 18 |

| Number of Observations |
|-----------------------------|
| Number of Observations Read |

| Covariance<br>Parameter<br>Estimates | Estimate | 0.02465 |
|--------------------------------------|----------|----------|
| Covar<br>Paran<br>Estin | Cov Parm | Residual |

| | 9.01 | 12.6 | 13.1 | 13.0 |
|---|---|---|---|---|
| Fit Statistics | -2 Res Log Likelihood | AIC (Smaller is Better) | AICC (Smaller is Better) | BIC (Smaller is Better) |

| | | | | Solution for Fixed Effects | for | Fixed Ef | fects | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | GRP | Estimate | Standard | DF | t Value | Pr > t | Alpha | Lower | Upper |
| Intercept | | | 5.3757 | 0.3995 | 11 | 13.45 | 1000.> | 0.05 | 4.4963 | 6.2551 |
| GRP | | 1 | 0.4928 | 0.1682 | 11 | 2.93 | 0.0137 | 0.05 | 0.1225 | 0.8631 |
| GRP | | 2 | -0.03700 | 0.1771 | 11 | -0.21 | 0.8383 | 0.05 | -0.4267 | 0.3527 |
| GRP | | 3 | 0.3271 | 0.2036 | 11 | 1.61 | 0.1364 | 0.05 | -0.1209 | 0.7752 |
| GRP | | 4 | 0 | | | | | | | |
| SEX | Ĺτι | | 0.1597 | 0.09566 | 11 | 1.67 | 0.1233 | 0.05 | -0.05088 | 0.3702 |
| SEX | M | | 0 | | | | | | | |
| AGE | | | 0.000470 | 0.000470 0.006104 | 11 | 0.08 | 0.9400 | 0.05 | -0.01297 | 0.01391 |
| BLWEIGHT | | | 0.001500 | 0.002900 | 11 | 0.52 | 0.6152 | 0.05 | -0.00488 | 0.007883 |

| בי ני | _ | Pr > F | _ | | |
|-------------|---------|--------|------|------|----------|
| | F Value | 11.55 | 2.79 | 10.0 | 0.27 |
| 5 | Den | 11 | 11 | 11 | 11 |
| ב<br>ה<br>ה | Num | 3 | 1 | Τ | 1 |
| 1750 | Effect | GRP | SEX | AGE | BLWEIGHT |

| | | Ä | stim | Estimates | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Standard | DF | t Value | ndard<br>Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| Mild vs Normal | -0.5298 | -0.5298 0.09573 11 -5.53 0.0002 0.1 -0.7017 -0.3579 | 11 | -5.53 | 0.0002 | 0.1 | -0.7017 | -0.3579 |
| Moderate vs Normal | -0.1657 | | 11 | -1.28 | 0.1292 11 -1.28 0.2262 0.1 -0.3977 0.06642 | 0.1 | -0.3977 | 0.06642 |
| Severe vs Normal | -0.4928 | | 11 | -2.93 | 0.1682 11 -2.93 0.0137 0.1 -0.7949 -0.1907 | 0.1 | -0.7949 | -0.1907 |

| | | | Leas | st S | Least Squares Means | ans | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect GRP | GRP | Estimate | Standard | DF | t Value | ndard Error DF t Value Pr > t Alpha | Alpha | Lower | Upper |
| GRP | 1 | 6.1083 | 6.1083 0.05215 11 117.12 | 11 | 117.12 | | 0.05 | ш, | 6.2231 |
| GRP | 2 | 5.5785 | 0.08611 11 | 11 | 64.78 | | 0.05 | <.0001 0.05 5.3889 5.7680 | 5.7680 |
| GRP | 3 | 5.9426 | 0.1273 11 | 11 | 46.70 | | 0.05 | <.0001 0.05 5.6625 6.2227 | 6.2227 |
| GRP | 4 | 5.6155 | 0.1657 11 | 11 | 33.89 | <.0001 | 0.05 | <.0001 0.05 5.2508 5.9801 | 5.9801 |

Supporting Document for Tables 15.4.3.5.1

The Mixed Procedure

ANAL=Additional Model 4 ANALYTEN=1 ANALYTE=Tepotinib PARM=AUCO-t (ng\*h/mL) PARAMCD=AUCLST

| Model Information | no |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| el<br>on | Values | F M |
|--------------------------|--------|-----|
| lass Level<br>nformation | Levels | 2 |
| υÄ | Class | SEX |

| | Τ | 9 | 0 | Τ | 18 |
|---|---|---|---|---|---|
| Dimensions | Covariance Parameters | Columns in X | Columns in Z | Subjects | Max Obs per Subject |

| Number of Observations | |
|-----------------------------|----|
| Number of Observations Read | 18 |
| Number of Observations Used | 18 |

Number of Observations

Number of Observations Not Used 0

| | | _ |
|--------------------------------------|----------|----------|
| Covariance<br>Parameter<br>Estimates | Estimate | 0.1263 |
| Covar<br>Parar<br>Estir | Cov Parm | Residual |

| Statistics | lhood 30.7 | Setter) 32.7 | Better) 33.1 | Better) 33.3 |
|---|---|---|---|---|
| Fit Statis | -2 Res Log Likelihood | AIC (Smaller is Better | AICC (Smaller is Be | BIC (Smaller is Bet |

| | | | Solution | n fo | Solution for Fixed Effects | Effects | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | Estimate | Standard | DF | t Value | t Value Pr > t | Alpha | ломот | Upper |
| Intercept | | 8.4293 | 0.9121 | 13 | 9.24 | <.0001 | 90.0 | 6.4587 | 10.3998 |
| XB | | -0.1272 | 0.1391 | 13 | -0.91 | 0.3771 | 0.05 | -0.4279 | 0.1734 |
| SEX | F | 0.2363 | 0.2142 | 13 | 1.10 | 0.2901 | 0.05 | -0.2265 | 0.6991 |
| SEX | М | 0 | | | | | | | |
| AGE | | 0.02223 | 0.01238 | 13 | 1.80 | 0.0958 | 0.05 | 0.05 -0.00451 | 0.04897 |
| BLWEIGHT | | -0.00026 | -0.00026 0.006382 13 | 13 | -0.04 | 0.9680 | 0.05 | 0.05 -0.01405 0.01353 | 0.01353 |

| Pr > F | 0.3771 |
|---------|----------------------------|
| F Value | 0.84 |
| Den | 13 |
| Num | 1 |
| Effect | XB |
| | Num Den F Value Pr > |

| Effects | Pr > F | 0.2901 | 0.0958 | 0.9680 |
|----------|-----------|--------|--------|----------|
| Fixed Ef | F Value | 1.22 | 3.23 | 00.00 |
| g of | Den<br>DF | 13 | 13 | 13 |
| Tests | Num<br>DF | 1 | 1 | 1 |
| Type 3 | Effect | SEX | AGE | BLWEIGHT |

Supporting Document for Tables 15.4.3.5.1

The Mixed Procedure

ANAL=Additional Model 4 ANALYTEN=1 ANALYTE=Tepotinib PARM=AUC0-inf (ng\*h/mL) PARAMCD=AUCIFP

| Model information | TI. |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| el | Values | F M |
|----------------------------|--------|-----|
| Class Level<br>Information | Levels | 2 |
| Cl | Class | SEX |

| | Н | 9 | 0 | Н | 18 |
|---|---|---|---|---|---|
| | | | | | Ι |
| Dimensions | Covariance Parameters | Columns in X | Columns in Z | Subjects | Max Obs per Subject |

| Number of Observations | |
|-----------------------------|----|
| Number of Observations Read | 18 |
| Number of Observations Used | 18 |

Number of Observations

Number of Observations Not Used 0

| Covariance<br>Parameter<br>Estimates | Estimate | 0.1201 |
|--------------------------------------|----------|----------|
| Covar<br>Parar<br>Estin | Cov Parm | Residual |

| | 30.1 | 32.1 | 32.4 | 32.6 |
|---|---|---|---|---|
| Fit Statistics | -2 Res Log Likelihood | AIC (Smaller is Better) | AICC (Smaller is Better) | BIC (Smaller is Better) |

| | | | Solution | n fc | Solution for Fixed Effects | Effects | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | Estimate | Standard | DF | DF t Value | Pr > t Alpha | Alpha | Lower | Upper |
| Intercept | | 8.4720 | 0.8894 | 13 | 6.53 | <.0001 | 0.05 | 9.5505 | 10.3934 |
| XB | | -0.1238 | 0.1357 | 13 | 16.0- | 0.3780 | 0.05 | -0.4170 0.1693 | 0.1693 |
| SEX | 댼 | 0.2359 | 0.2089 | 13 | 1.13 | 0.2791 | | 0.05 -0.2154 | 0.6872 |
| SEX | М | 0 | | | | | | | |
| AGE | | 0.02181 | 0.01207 | 13 | 1.81 | 0.0939 | | 0.05 -0.00426 | 0.04788 |
| BLWEIGHT | | -0.00012 | -0.00012 0.006224 | 13 | -0.02 | 0.9849 | | 0.05 -0.01357 0.01333 | 0.01333 |

| Pr > F | 0848.0 |
|-----------|-----------------------|
| F Value | 0.83 |
| Den<br>DF | 13 |
| Num<br>DF | 1 |
| Effect | XB |
| | ffect DF F Value Pr > |

| Effects | Pr > F | 0.2791 | 0.0939 | 0.9849 |
|----------|---------|--------|--------|----------|
| Fixed Ef | F Value | 1.28 | 3.27 | 00.00 |
| 3 of | Den | 13 | 13 | 13 |
| Tests | Num | 1 | 1 | 1 |
| Type 3 | Effect | SEX | AGE | BLWEIGHT |

Supporting Document for Tables 15.4.3.5.1

The Mixed Procedure

ANAL=Additional Model 4 ANALYTEN=1 ANALYTE=Tepotinib PARM=Cmax (ng/mL) PARAMCD=CMAX

| Model Information | no |
|---------------------------|-------------|
| Data Set | WORK.PK |
| Dependent Variable | LNEST |
| Covariance Structure | Diagonal |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Model-Based |
| Degrees of Freedom Method | Residual |

| el<br>on | Values | F M |
|--------------------------|--------|-----|
| lass Level<br>nformation | Levels | 2 |
| บี่ | Class | SEX |

| Dimensions | |
|-----------------------|----|
| Covariance Parameters | 1 |
| Columns in X | 9 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs per Subject | 18 |

| Number of Observations | |
|-----------------------------|----|
| Number of Observations Read | 18 |
| Number of Observations Used | 18 |

Number of Observations
Number of Observations Not Used

| | ۵) | 9 |
|--------------------------------------|----------|----------|
| covariance<br>Parameter<br>Estimates | Estimate | 95720.0 |
| Covar<br>Parar<br>Estir | Cov Parm | Residual |

| Fit Statistics -2 Res Log Likelihood AIC (Smaller is Better) | 20.5 |
|--------------------------------------------------------------|------|
| AICC (Smaller is Better) | 22.9 |
| BIC (Smaller is Better) | 23.1 |

| | | | Solutio | on f | Solution for Fixed Effects | Effects | | | |
|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | Estimate | Standard<br>Error | DF | t Value | t Value $ Pr > t $ Alpha | Alpha | Lower | Upper |
| Intercept | | 4.6364 | 0.6158 | 13 | 7.53 | <.0001 | 90.0 | 3.3061 | 5.9667 |
| XB | | -0.2404 | -0.2404 0.09394 13 | 13 | -2.56 | 0.0238 | 0.05 | | -0.4433 -0.03746 |
| SEX | F | 0.1546 | 0.1446 13 | 13 | 1.07 | 0.3044 | 0.05 | -0.1578 | 0.4671 |
| SEX | М | 0 | | | | | | | |
| AGE | | 0.009421 | 0.008355 | 13 | 1.13 | 0.2799 | 0.05 | 0.05 -0.00863 | 0.02747 |
| BLWEIGHT | | 0.000026 | 0.000026 0.004309 | 13 | 0.01 | 0.9952 | | 0.05 -0.00928 0.009334 | 0.009334 |

| | _ | |
|-------|-----------|------|
| Ω | | 0238 |
| Ĺ. | Pr | 0.0 |
| Effec | | 2 |
| <br>О | Value | 6.5 |
| Fixe | F | |
| oĘ | Den<br>DF | 13 |
| Tests | Num | 1 |
| m | | |
| Type | Effect | XB |

| Effects | Pr > F | 0.3044 | 0.2799 | 0.9952 |
|----------|-----------|--------|--------|----------|
| Fixed Ef | F Value | 1.14 | 1.27 | 00.00 |
| s of | Den<br>DF | 13 | 13 | 13 |
| Tests | Num<br>DF | 1 | 1 | 1 |
| Type 3 | Effect | SEX | AGE | BLWEIGHT |